

## A PHASE 4, OPEN-LABEL, SINGLE-ARM, MULTICENTER STUDY TO DESCRIBE THE SAFETY OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN ADULTS 18 TO 49 YEARS OF AGE IN INDIA

**Study Intervention Number:** PF-05208760

Study Intervention Name: 13-valent Pneumococcal Conjugate Vaccine

US IND Number: N/A
EudraCT Number: N/A
ClinicalTrials.gov ID: TBD

**Protocol Number:** B1851214

Phase: 4

Brief Title: A Phase 4 Safety Study of 13vPnC in Adults 18 to 49 Years of Age in India



# **Document History**

| Document | Version Date |
|-------------------|-----------------|
| Original protocol | 15 October 2021 |

# TABLE OF CONTENTS

| LIST OF TABLES | 7 |
|---|---|
| 1. PROTOCOL SUMMARY | 8 |
| 1.1. Synopsis | 8 |
| 1.2. Schema. | 10 |
| 1.3. Schedule of Activities | 10 |
| 2. INTRODUCTION | 11 |
| 2.1. Study Rationale | 13 |
| 2.2. Background | 13 |
| 2.3. Benefit/Risk Assessment | 14 |
| 2.3.1. Risk Assessment | 15 |
| 2.3.2. Benefit Assessment | 16 |
| 2.3.3. Overall Benefit/Risk Conclusion | 16 |
| 3. OBJECTIVES, ENDPOINTS, AND ESTIMANDS | 16 |
| 4. STUDY DESIGN | 16 |
| 4.1. Overall Design | 16 |
| 4.2. Scientific Rationale for Study Design | 16 |
| 4.3. Justification for Dose | 17 |
| 4.4. End of Study Definition | 17 |
| 5. STUDY POPULATION | 17 |
| 5.1. Inclusion Criteria | 17 |
| 5.2. Exclusion Criteria | 18 |
| 5.3. Lifestyle Considerations | 19 |
| 5.3.1. Contraception | 19 |
| 5.4. Screen Failures | 19 |
| 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Administration of Study Intervention | 20 |
| 5.5.1. Temporary Delay Criteria | 20 |
| 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY | 20 |
| 6.1. Study Intervention(s) Administered | |
| 6.1.1. Administration | 20 |
| 6.1.2. Medical Devices | 21 |

| 6.2. Preparation, Handling, Storage, and Accountability | 21 |
|---|---|
| 6.2.1. Preparation and Dispensing | 22 |
| 6.3. Measures to Minimize Bias: Randomization and Blinding | 22 |
| 6.3.1. Allocation to Study Intervention | 22 |
| 6.4. Study Intervention Compliance | 22 |
| 6.5. Dose Modification | 22 |
| 6.6. Continued Access to Study Intervention After the End of the Study | 22 |
| 6.7. Treatment of Overdose | 23 |
| 6.8. Concomitant Therapy | 23 |
| 6.8.1. Prohibited During the Study | 23 |
| 6.8.2. Permitted During the Study | 23 |
| 6.8.3. Recording Prior and Concomitant Vaccines and Concomitant Treatments | 24 |
| 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL | 24 |
| 7.1. Discontinuation of Study Intervention. | 24 |
| 7.1.1. Participant Discontinuation/Withdrawal From the Study | 24 |
| 7.1.2. Withdrawal of Consent | |
| 7.2. Lost to Follow-Up | 25 |
| 8. STUDY ASSESSMENTS AND PROCEDURES | 25 |
| 8.1. Efficacy and/or Immunogenicity Assessments | 26 |
| 8.2. Safety Assessments | 26 |
| 8.2.1. Physical Examinations | 27 |
| 8.2.2. Participant Electronic Diary | 27 |
| 8.2.3. Grading Scale for Prompted Events | 27 |
| 8.2.3.1. Local Reactions | 28 |
| 8.2.3.2. Systemic Events – Systemic Symptoms and Fever | 29 |
| 8.2.4. Clinical Safety Laboratory Assessments | 30 |
| 8.2.5. Pregnancy Testing | 30 |
| 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting | 30 |
| 8.3.1. Time Period and Frequency for Collecting AE and SAE Information | 31 |
| 8.3.1.1. Reporting SAEs to Pfizer Safety | 31 |

| 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF | 32 |
|---|---|
| 8.3.2. Method of Detecting AEs and SAEs | 32 |
| 8.3.3. Follow-Up of AEs and SAEs | 32 |
| 8.3.4. Regulatory Reporting Requirements for SAEs | 32 |
| 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure | 33 |
| 8.3.5.1. Exposure During Pregnancy | 33 |
| 8.3.5.2. Exposure During Breastfeeding | 34 |
| 8.3.5.3. Occupational Exposure | 35 |
| 8.3.6. Cardiovascular and Death Events | 35 |
| 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs | 35 |
| 8.3.8. Adverse Events of Special Interest | 35 |
| 8.3.8.1. Lack of Efficacy | 35 |
| 8.3.9. Medical Device Deficiencies | 36 |
| 8.3.9.1. Time Period for Detecting Medical Device Deficiencies | 36 |
| 8.3.9.2. Follow-Up of Medical Device Deficiencies | 36 |
| 8.3.9.3. Prompt Reporting of Device Deficiencies to the Sponsor | 36 |
| 8.3.9.4. Regulatory Reporting Requirements for Device Deficiencies | 37 |
| 8.3.10. Medication Errors | 37 |
| 8.4. Pharmacokinetics | 38 |
| 8.5. Genetics | 38 |
| 8.5.1. Specified Genetics | 38 |
| 8.6. Biomarkers | 38 |
| 8.7. Immunogenicity Assessments | 38 |
| 8.8. Health Economics | 38 |
| 8.9. Study Procedures | 39 |
| 8.9.1. Visit 1 (Vaccination 1 – Day 1) | 39 |
| 8.9.2. Visit 2 (Follow-Up – 28 to 42 Days After Vaccination 1 [Study Days 29 to 43]) | 41 |
| 8.10. Unscheduled Visits | 41 |
| 9. STATISTICAL CONSIDERATIONS | 42 |

| 9.1. Statistical Hypotheses | 42 |
|---|---|
| 9.1.1. Estimands | 42 |
| 9.2. Analysis Sets. | 43 |
| 9.3. Statistical Analyses | 43 |
| 9.3.1. General Considerations | 43 |
| 9.3.2. Analysis for Binary Data | 43 |
| 9.3.3. Analysis for Continuous Data | 43 |
| 9.3.4. Primary Endpoint(s)/Estimand(s) Analysis | 44 |
| 9.4. Interim Analyses | 44 |
| 9.5. Sample Size Determination | 44 |
| 10. SUPPORTING DOCUMENTATION AND OPERATIONAL | |
| CONSIDERATIONS | 45 |
| 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations | 45 |
| 10.1.1. Regulatory and Ethical Considerations | 45 |
| 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 45 |
| 10.1.2. Financial Disclosure | 46 |
| 10.1.3. Informed Consent Process | 46 |
| 10.1.4. Data Protection | 47 |
| 10.1.5. Committees Structure | 47 |
| CCI | |
| 10.1.6. Dissemination of Clinical Study Data | 47 |
| 10.1.7. Data Quality Assurance | 49 |
| 10.1.8. Source Documents | 50 |
| 10.1.9. Study and Site Start and Closure | 50 |
| 10.1.10. Publication Policy | 51 |
| 10.1.11. Sponsor's Qualified Medical Personnel | 52 |
| 10.2. Appendix 2: Clinical Laboratory Tests | 53 |
| 10.3. Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting | 54 |
| 10.3.1. Definition of AE | 54 |
| 10.3.2. Definition of an SAE | 55 |

| 10 | 0.3.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period | 57 |
|---|---|---|
| 1/ | | |
| | 0.3.4. Reporting of SAEs | |
| | ppendix 4: Contraceptive and Barrier Guidance | |
| | 0.4.1. Male Participant Reproductive Inclusion Criteria | |
| | 0.4.2. Female Participant Reproductive Inclusion Criteria | |
| 10 | 0.4.3. Woman of Childbearing Potential | 63 |
| 10 | 0.4.4. Contraception Methods | 64 |
| | ppendix 5: Liver Safety: Suggested Actions and Follow-Up Assessments ntial Cases of Drug-Induced Liver Injury | 66 |
| Defi | ppendix 6: AEs, ADEs, SAEs, SADEs, USADEs, and Device ciencies: Definitions and Procedures for Recording, Evaluating, ow-Up, and Reporting in Medical Device Studies | 68 |
| 10 | 0.6.1. Definition of AE and ADE | 68 |
| 10 | 0.6.2. Definition of SAE, SADE, and USADE | 68 |
| 10 | 0.6.3. Definition of Device Deficiency | 69 |
| 10 | 0.6.4. Recording/Reporting and Follow-Up of Medical Device Deficiencies | 69 |
| 1( | 0.6.5. Reporting of SAEs | |
| | 0.6.6. Reporting of SADEs | |
| | ppendix 7: Alternative Measures During Public Emergencies | |
| | 0.7.1. Telehealth Visits | |
| | ppendix 8: Abbreviations | |
| | NCES | |
| | LIST OF TABLES | |
| Table 1. | Grading Scales for Local Reactions | 28 |
| Table 2. | Grading Scales for Systemic Events | 29 |
| Table 3. | Ranges for Fever | |
| Table 4. | Probability of Detecting at Least 1 AE | |

#### 1. PROTOCOL SUMMARY

## 1.1. Synopsis

Streptococcus pneumoniae is a significant cause of invasive disease (sepsis, meningitis) and pneumonia globally in adults. Elderly adults or those with certain underlying medical conditions or who smoke are at increased risk for developing severe pneumococcal disease and its complications. The risk in adults with multiple underlying conditions can approach or exceed that of the elderly in some cases. Furthermore, the treatment of pneumococcal infections is becoming more difficult because of the increased prevalence of antibiotic-resistant *S pneumoniae* strains.

The 13-valent pneumococcal conjugate vaccine (13vPnC; Prevenar 13®) is a pneumococcal conjugate vaccine that contains the capsular polysaccharides of 13 different pneumococcal serotypes, each individually conjugated to a protein carrier (CRM<sub>197</sub>), a nontoxic variant of diphtheria toxin. In contrast to the other type of pneumococcal vaccine used in adults, the 23-valent pneumococcal polysaccharide vaccine (PPSV23) containing unconjugated polysaccharides, 13vPnC elicits a T-cell–dependent immune response. T cells provide the signals required for the generation of B-cell memory. 13vPnC therefore has the potential for eliciting a memory response on subsequent natural exposure. Additionally, 13vPnC has demonstrated efficacy against VT pneumonia and IPD in a randomized efficacy trial and in real-world effectiveness trials.

13vPnC has been approved for use in adults since 2011, initially licensed for adults 50 years of age and subsequently in 2016 (US) and 2015 (Europe) for adults 18 years of age and older in the US, Europe, and other countries, for the prevention of VT pneumococcal disease. Licensure was based on demonstration of immune responses that were comparable to, or better than, PPSV23 responses, and subsequently 13vPnC demonstrated efficacy against CAP and IPD due to 13vPnC serotypes in a randomized, controlled efficacy trial in adults 65 years of age and older.

Safety and immunogenicity data generated with 13vPnC in India in pediatric populations (6 weeks to 17 years of age) and adults over 50 years of age have shown that the clinical findings with 13vPnC in Indian populations are consistent with global data. These data have supported 13vPnC licensure and indications for use in these age groups in India. The data from India generated in all other age groups and the global data with 13vPnC specifically in adults 18 to 49 years of age, showing acceptable safety and robust immunogenicity in that age group, support a conclusion that 13vPnC will also be safe and immunogenic in the Indian population of adults 18 to 49 years of age. The DCGI granted approval for this age group in May 2021.

This study, B1851214, in the Indian population of adults 18 to 49 years of age is being conducted based on SEC recommendation and the condition mentioned in the DCGI approval to conduct a Phase 4 clinical trial. This protocol describes the study to meet that commitment. In this study, safety data will be collected in adults 18 to 49 years of age. E-diaries will be given to the participants to report local reactions and systemic events for

7 days after vaccination. Investigators will collect other AEs at the follow-up visit 1 month after vaccination.

#### STUDY OBJECTIVES, ENDPOINTS, AND ESTIMANDS

| Objective | Objective Endpoints Estimands | |
|---|---|---|
| Primary: | Primary: | Primary: |
| To describe the safety profile of 13vPnC when administered to adults 18 to 49 years of age | <ul> <li>Prompted local reactions (redness, swelling, and pain at the injection site)</li> <li>Prompted systemic events (fever, headache, fatigue, muscle pain, and joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> | In participants receiving the single dose of study intervention and having safety follow-up after vaccination, the percentage of participants reporting: • Prompted local reactions within 7 days after vaccination • Prompted systemic events within 7 days after vaccination • AEs within 1 month after vaccination • SAEs within 1 month after vaccination |

#### STUDY DESIGN

This is a Phase 4, open-label, single-arm, multicenter study in which participants 18 to 49 years of age will receive a single intramuscular administration of 13vPnC. This study will be conducted in India.

## **Intervention Groups and Duration**

Each participant will participate in the study for approximately 1 month. Based on an estimated enrollment timing, the study duration will be approximately 5 months.

## **Number of Participants**

Approximately 200 participants will be vaccinated.



#### **Statistical Methods**

There is no formal hypothesis test for any safety results. All statistical analyses will be descriptive.

The primary safety objective will be evaluated by descriptive summary statistics (including counts and percentages of participants and the associated 2-sided 95% CIs) for local reactions at the injection site, systemic events, AEs, and SAEs for the entire cohort. With 200 vaccinated participants, the study will provide a greater than 86% chance of observing at least 1 AE if the true rate is at least 1%.

#### 1.2. Schema

Not applicable.

#### 1.3. Schedule of Activities

The SoA table provides an overview of the protocol visits and procedures. Refer to the STUDY ASSESSMENTS AND PROCEDURES section of the protocol for detailed information on each procedure and assessment required for compliance with the protocol.

The investigator may schedule visits (unplanned visits) in addition to those listed in the SoA table, in order to conduct evaluations or assessments required to protect the well-being of the participant.

| Visit Number | 1 | 2 |
|---|---|---|
| Visit ID | Vaccination | Follow-Up<br>Visit |
| Visit Window (Days) | Day 1 | 28 to 42 Days<br>After Visit 1 |
| Visit Type | Clinic Visit | Clinic Visit |
| Informed consent | X | |
| Assign participant number via the IRT | X | |
| Record demography | X | |
| Perform clinical assessment, including medical history | X | |
| Perform a clinical assessment, if appropriate | | X |
| Perform pregnancy test, if applicable | X | |
| Record nonstudy vaccinations | X | X |
| Obtain prevaccination oral temperature | X | |
| Contraception check, if applicable | X | |
| Review inclusion and exclusion criteria | X | |
| Review temporary delay criteria | X | |
| Administer study intervention | X | |
| Observe and record acute reactions for 20 minutes after 13vPnC administration | X | |
| Provide participant with an e-diary (device or application, if used), digital thermometer, and measuring device and instruct to collect prompted local reactions, and systemic events for 7 days after vaccination | X | |
| Provide a participant contact card | X | |
| Review e-diary data (daily is optimal during 7-day diary period) | X | X |
| Review reactogenicity e-diary symptoms with participant and obtain stop dates where applicable | | X |
| Collect e-diary or assist the participant to delete the application, if applicable | | X |
| AEs and SAEs collection | X | X |

Abbreviation: IRT = interactive response technology.

#### 2. INTRODUCTION

#### **Indication of 13vPnC in India**

Prevenar 13 (13vPnC) is currently approved in India for the following indications:

For active immunization for the prevention of disease caused by *S pneumoniae* serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F (including sepsis, meningitis, bacteremia, pneumonia, and AOM) in infants and children 6 weeks to 5 years of age.

For active immunization for prevention of pneumonia and invasive disease caused by *S pneumoniae* serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F in children 6 to 17 years of age.

For active immunization for the prevention of pneumonia and invasive disease caused by *S pneumoniae* serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F in adults 18 to 49 years of age.

For active immunization for the prevention of pneumonia and invasive disease caused by *S pneumoniae* serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F in adults 50 years of age and older.

#### **Pneumococcal Disease**

## Pneumococcal Disease Burden

S pneumoniae are gram-positive encapsulated cocci that are a leading cause of bacteremia, bacterial meningitis, pneumonia, and AOM and continue to be a major global public health concern. Serious pneumococcal disease may occur at any age; however, children <5 years and adults ≥65 years of age are at particularly increased risk.¹ Individuals with certain comorbidities and immunocompromising conditions are also at risk, especially persons with chronic heart, lung, liver, and renal disease, as well as those who are functionally asplenic. Among nonelderly immunocompetent individuals, cigarette smoking is considered the strongest independent risk factor for IPD.²

In India, *S pneumoniae* is associated with high disease burden and mortality among young children.<sup>3</sup> Pneumococcal pneumonia is the most common clinical presentation of pneumococcal disease among adults. Adults with certain medical conditions are at highest risk for IPD. Conditions that place adults at highest risk for IPD include immunosuppressive conditions from disease or drugs, functional or anatomic asplenia, and renal disease. Other conditions that increase the risk of IPD in adults include chronic heart disease, lung disease (including asthma), liver disease, smoking cigarettes, alcoholism, CSF leak, and having a cochlear implant.<sup>4</sup>

Several studies from India have documented the burden of pneumococcal disease, both IPD and pneumonia, in the adult population >18 years of age. <sup>5,6</sup> Across various studies that have identified the etiology of CAP in adults in India, *S pneumoniae* has been the most commonly identified pathogen, accounting for about 32% to 55% of cases. <sup>7,8,9,10</sup>

Various Indian medical societies, such as the Indian Society of Nephrology, Indian Medical Association, Indian Chest Society, and Indian Association of Occupational Health, recommend 13vPnC for adults, including those in the 18- to 49-year age group. 11,12,13,14

## Vaccines to Prevent Pneumococcal Disease

The polysaccharide capsule has been identified as an important virulence factor for this pathogen. While more than 95 pneumococcal serotypes, differentiated by their capsular polysaccharide composition, have been identified, serious disease is generally caused by a smaller subset of serotypes. <sup>15,16</sup> Anticapsular antibodies directed against the specific serotype bind to the capsule and promote complement-mediated opsonophagocytic killing and clearance of the organism. <sup>17</sup> Pneumococcal disease can be prevented with polysaccharide-based vaccines that induce antibody responses with functional (opsonophagocytic) activity and target the capsular serotypes responsible for disease. <sup>18</sup>

#### Pneumococcal Polysaccharide Vaccines

Vaccines containing free polysaccharides have been licensed since the 1970s. One such vaccine, PPSV23, has been licensed in the US since 1983. 19,20 PPSV23 contains capsular polysaccharides for 23 serotypes (1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, and 33F). Pneumococcal vaccines containing free polysaccharides, such as PPSV23, elicit a T-cell-independent immune response. Unconjugated polysaccharide vaccines do not induce robust responses in certain populations (eg, immunocompromised persons and children <2 years of age), nor do they generate immunologic memory, so their protective effect wanes over 2 to 5 years. 1,20,21,22 Moreover, their ability to prevent nonbacteremic pneumonia, CAP, and AOM is limited or lacking. 18,22,23,24,25 In addition, polysaccharide vaccines do not reduce VT nasopharyngeal carriage, which is important for herd immunity. PPSV23 is not recommended for children <2 years of age and is only recommended in children >2 years of age who are at high risk for IPD to provide some degree of protection from disease caused by serotypes not covered by existing pneumococcal conjugate vaccines.

## Pneumococcal Polysaccharide Conjugate Vaccines

Pneumococcal conjugate vaccines contain polysaccharides that are covalently linked (conjugated) to an immunogenic protein. This modification results in T-cell—dependent immune responses, which have been shown to be protective in young children, older adults, and populations with high-risk conditions. <sup>21,26</sup> 7vPnC was the first pneumococcal conjugate vaccine to be licensed (2000) and was indicated for prevention of pneumococcal disease in infants and young children on the basis of efficacy studies.

13vPnC was developed to expand serotype coverage beyond that of 7vPnC and was initially licensed in 2010 (US). 13vPnC includes the same *S pneumoniae* serotypes as 7vPnC and an additional 6 polysaccharide conjugates for serotypes 1, 3, 5, 6A, 7F, and 19A. <sup>26,27,28</sup> The vaccine was initially licensed for use in infants and young children based on comparisons of serotype-specific serum IgG antibody concentrations to 7vPnC, with supportive data to demonstrate the functional activity of the immune responses. 13vPnC has also been licensed in adults based on demonstration of comparable or higher levels of functional (opsonophagocytic) antibodies compared to PPSV23 and subsequently was shown to be efficacious against VT CAP and IPD in the randomized, placebo-controlled study of approximately 84,000 adults 65 years of age and older (CAPiTA study). <sup>29</sup> 13vPnC was licensed for populations 18 to 59 years of age by showing that immune responses elicited in that population were comparable to, or higher than, responses in the older age groups where efficacy was previously demonstrated. Following the introduction of 13vPnC, real-world vaccine effectiveness has been observed against 13vPnC-type IPD and CAP in vaccinated populations. <sup>30</sup>

#### 2.1. Study Rationale

In India, 13vPnC has been clinically evaluated and demonstrated to be safe and immunogenic in Indian infants, children, adolescents, and adults 50 years of age and above. The vaccine was approved in infants and children 6 weeks to 5 years of age, in adults 50 years of age and older, and in children 6 to 17 years of age.

The safety and immunogenicity findings generated in India in infants, children through adolescents, and adults 50 years of age and older are generally consistent with data generated from global studies in these populations. Based on the favorable findings in the pediatric and older adult studies with 13vPnC in India, as well as the global data in adults 18 to 49 years of age, showing that 13vPnC has an acceptable safety profile and elicits robust immune responses for all 13 serotypes, the DCGI granted approval for this age group in May 2021.

This study, B1851214, in the Indian population 18 to 49 years of age is being conducted based on SEC recommendation and the condition mentioned in DCGI approval to conduct a Phase 4 clinical trial. This protocol describes the study to meet that commitment.

In this study, safety data will be collected in adults 18 to 49 years of age. E-diaries will be given to the participants to report local reactions and systemic events for 7 days after vaccination. Investigators will collect other AEs at the follow-up visit 1 month after vaccination.

## 2.2. Background

This study is designed to meet a commitment to obtain safety data for 13vPnC in the 18- to 49-year-old population in India, where 13vPnC was granted an indication by the DCGI in May 2021.

The study will evaluate the safety of 13vPnC given as a single dose according to the posology in the approved label. The safety assessments to be performed are based on prior studies of 13vPnC in adults and adolescents in India.

This study is defined as a PASS and is being conducted at the request of the DCGI.

#### 2.3. Benefit/Risk Assessment

More detailed information about the known and expected benefits and risks and reasonably expected AEs of 13vPnC may be found in the Indian Prevenar 13 (13vPnC) package insert, which is the SRSD for this study.

## 2.3.1. Risk Assessment

| Potential Risk of Clinical Significance | Summary of Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| | Study Intervention(s): 13vPnC | |
| The relevant key risks associated with 13vPnC include: local reactions (injection site pain, redness, and swelling); systemic events (fever, headache, fatigue, joint pain, and muscle pain); and allergic reactions, including skin rash, facial edema, | The risks are based on the Indian Prevenar 13 (13vPnC) package insert for adults in this age group. | Eligibility criteria have been selected to ensure that only appropriate participants are included in the study (see Section 5). E-diary and AE data will be monitored by the investigator (or designee) and sponsor. |
| bronchospasm, shortness of breath, or severe allergic reaction (eg, anaphylactic shock). | | All study participants will be observed for 20 minutes after vaccination. |
| | Other | |
| The COVID-19 pandemic may pose risks to study participation. | Participants may have increased risk of SARS-CoV-2 infection by undergoing a study procedure at a study facility. | Pfizer will work with sites to ensure an appropriate COVID-19 prevention strategy. |

#### 2.3.2. Benefit Assessment

13vPnC is anticipated to provide a benefit to a participant in the prevention of pneumonia and invasive disease caused by vaccine serotypes.

#### 2.3.3. Overall Benefit/Risk Conclusion

Taking into account the measures to minimize risk to study participants, the potential risks identified in association with 13vPnC are justified by the anticipated benefits that may be afforded to participants.

#### 3. OBJECTIVES, ENDPOINTS, AND ESTIMANDS

| Objective | Endpoints | Estimands |
|---|---|---|
| Primary: | Primary: | Primary: |
| To describe the safety profile of 13vPnC when administered to adults 18 to 49 years of age | <ul> <li>Prompted local reactions (redness, swelling, and pain at the injection site)</li> <li>Prompted systemic events (fever, headache, fatigue, muscle pain, and joint pain)</li> <li>AEs</li> <li>SAEs</li> </ul> | In participants receiving the single dose of study intervention and having safety follow-up after vaccination, the percentage of participants reporting: • Prompted local reactions within 7 days after vaccination • Prompted systemic events within 7 days after vaccination • AEs within 1 month after vaccination • SAEs within 1 month after vaccination |

#### 4. STUDY DESIGN

#### 4.1. Overall Design

This is a Phase 4, open-label, single-arm, multicenter study in which approximately 200 adults 18 to 49 years of age will receive 1 intramuscular dose of 13vPnC. This study will be conducted in India. Participants will take part in the study for approximately 1 month.

Based on an estimated enrollment period of 4 months, the total study duration will be approximately 5 months.

## 4.2. Scientific Rationale for Study Design

This protocol is being conducted at the request of the DCGI and will obtain safety data in the 18- to 49-year-old population in India, where 13vPnC was granted an indication by the DCGI in May 2021.

The study will evaluate the safety of 13vPnC given as a single dose according to the posology in the approved label. The safety assessments to be performed are based on prior studies of 13vPnC in adults and adolescents in India.

#### 4.3. Justification for Dose

The study follows the dosing indicated for this age group in the Indian Prevenar 13 (13vPnC) package insert.

For this device, the term "dose" refers to administration of vaccine.

#### 4.4. End of Study Definition

The end of the study is defined as the date of the last visit of the last participant in the study.

#### 5. STUDY POPULATION

This study can fulfill its objective only if appropriate participants are enrolled. The following eligibility criteria are designed to select participants for whom participation in the study is considered appropriate. All relevant medical and nonmedical conditions should be taken into consideration when deciding whether a particular participant is suitable for this protocol.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1. Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

### Age and Sex:

- 1. Generally healthy participants between the ages of  $\geq$ 18 and <50 years, at Visit 1.
  - Refer to Appendix 4 for reproductive criteria for male (Section 10.4.1) and female (Section 10.4.2) participants.

#### **Type of Participant and Disease Characteristics:**

- 2. Participants who are willing and able to comply with all scheduled visits, treatment plan, lifestyle considerations, and other study procedures.
- 3. Participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

Note: Participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 12 weeks before enrollment, can be included.

#### **Informed Consent:**

4. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

#### 5.2. Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### **Medical Conditions:**

- 1. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of 13vPnC, or to any other diphtheria toxoid—containing vaccine.
- 2. History of microbiologically-proven invasive disease caused by *S pneumoniae*.
- 3. Known or suspected immune deficiency or suppression.
- 4. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
- 5. Congenital, functional, or surgical asplenia.
- 6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

## **Prior/Concomitant Therapy:**

- 7. Previous vaccination with any pneumococcal vaccine, or planned receipt of any pneumococcal vaccine through study participation.
- 8. Currently receives treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, or planned receipt during the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intraarticular, intrabursal, or topical (skin, eyes, or ears) corticosteroids are permitted.
- 9. Receipt of blood/plasma products or immunoglobulin within the 60 days before study intervention administration, or planned receipt during the study.

## **Prior/Concurrent Clinical Study Experience:**

10. Participation in other studies involving investigational drugs, investigational vaccines (with the exception of vaccines authorized by the DCGI for pandemic use), or investigational devices within 28 days prior to study entry and/or during study participation. Participation in purely observational studies is acceptable.

#### **Diagnostic Assessments:**

Not applicable.

#### **Other Exclusions:**

11. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

## 5.3. Lifestyle Considerations

## 5.3.1. Contraception

The investigator or his or her designee, in consultation with the participant, will confirm that the participant has selected an appropriate method of contraception for the individual participant and his or her partner(s) from the permitted list of contraception methods (see Appendix 4, Section 10.4.4) and will confirm that the participant has been instructed in its consistent and correct use. At time points indicated in the SoA, the investigator or designee will inform the participant of the need to use acceptable/highly effective contraception consistently and correctly and document the conversation and the participant's affirmation in the participant's chart (participants need to affirm their consistent and correct use of at least 1 of the selected methods of contraception) considering that their risk for pregnancy may have changed since the last visit. In addition, the investigator or designee will instruct the participant to call immediately if the selected contraception method is discontinued or if pregnancy is known or suspected in the participant or partner.

#### 5.4. Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently enrolled in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the CONSORT publishing requirements and to respond to queries from regulatory authorities. Minimal information includes demography, screen failure details, eligibility criteria, and any SAE.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be rescreened.

# 5.5. Criteria for Temporarily Delaying Enrollment/Randomization/Administration of Study Intervention

The following conditions may allow a participant to be vaccinated once the conditions have resolved and the participant is otherwise eligible:

## 5.5.1. Temporary Delay Criteria

The following conditions are temporary or self-limiting and a participant may be vaccinated in the study once the condition(s) has/have resolved and no other exclusion criteria are met.

- Current febrile illness (body temperature ≥100.4°F [≥38.0°C]) or other acute illness within 48 hours before study intervention administration.
- Receipt of any inactivated or otherwise nonlive vaccine within 14 days or any live vaccine within 28 days before study intervention administration.

## 6. STUDY INTERVENTION(S) AND CONCOMITANT THERAPY

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, medical device(s), or study procedure(s) intended to be administered to a study participant according to the study protocol.

For the purposes of this protocol, 13vPnC may be used synonymously with study intervention.

#### 6.1. Study Intervention(s) Administered

13vPnC contains saccharides from pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F individually conjugated to nontoxic diphtheria toxin CRM<sub>197</sub>. The vaccine is formulated to contain 2.2 μg of each saccharide, except for 4.4 μg of 6B, per 0.5-mL dose. The vaccine contains 5 mM succinate buffer, 0.85% sodium chloride, 0.02% polysorbate 80, and 0.125 mg aluminum as aluminum phosphate, per 0.5-mL dose.

13vPnC will be provided as a 0.5-mL dose in a prefilled syringe.

#### 6.1.1. Administration

At Visit 1, all participants will receive a single dose (0.5 mL) of 13vPnC intramuscularly into the deltoid muscle.

Standard vaccination practices must be observed and vaccine must not be injected into blood vessels. Appropriate medication and other supportive measures for management of an acute hypersensitivity reaction should be available in accordance with local guidelines for standard immunization practices.

Administration of study interventions should be performed by an appropriately qualified, GCP-trained, and vaccine-experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacist, or medical assistant) as allowed by local, state, and institutional guidance.

Study intervention administration details will be recorded on the CRF.

#### **6.1.2.** Medical Devices

In this study, medical devices being deployed are the prefilled syringes containing 13vPnC. Instructions for medical device use are provided in the IP manual or in the package insert.

Medical device incidents, including those resulting from malfunctions of the device, must be detected, documented, and reported by the unblinded study personnel throughout the study. Please refer to Section 8.3.9 and Section 10.6 for details.

## 6.2. Preparation, Handling, Storage, and Accountability

1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study interventions received and any discrepancies are reported and resolved before use of the study intervention.





Upon identification of a product complaint, notify the sponsor within 1 business day of discovery as described in the IP manual.

## 6.2.1. Preparation and Dispensing

See the IP manual, package insert, or equivalent for instructions on how to prepare the study intervention for administration. Study intervention should be prepared and dispensed by an appropriately qualified and experienced member of the study staff (eg, physician, nurse, physician's assistant, nurse practitioner, pharmacy assistant/technician, or pharmacist) as allowed by local, state, and institutional guidance.

## 6.3. Measures to Minimize Bias: Randomization and Blinding

## 6.3.1. Allocation to Study Intervention

This is a Phase 4 single-arm, open-label study.

The study intervention will be dispensed at the study visits summarized in the SoA.

## **6.4. Study Intervention Compliance**

When participants are dosed at the site, they will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of each dose administered in the clinic will be recorded in the source documents and recorded in the CRF. The dose of study intervention and study participant ID will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention.

#### 6.5. Dose Modification

Not applicable.

#### 6.6. Continued Access to Study Intervention After the End of the Study

Not applicable.

#### 6.7. Treatment of Overdose

For this study, any dose of study intervention greater than 1 dose of study intervention within a 24-hour time period will be considered an overdose.

Pfizer does not recommend specific treatment for an overdose. In the event of an overdose, the investigator should:

- 1. Contact the medical monitor within 24 hours.
- 2. Closely monitor the participant for any AEs/SAEs.
- 3. Document the quantity of the excess dose as well as the duration of the overdose in the CRF.
- 4. Overdose is reportable to Pfizer Safety only when associated with an SAE.

## 6.8. Concomitant Therapy

## 6.8.1. Prohibited During the Study

- Receipt of any investigational vaccines, drugs, or medical devices is prohibited during study participation.
- Receipt of a nonstudy pneumococcal vaccine is prohibited during study participation.
- Receipt of any other licensed nonstudy vaccine is prohibited during the study, unless medically necessary.
- Receipt of blood/plasma products, immunoglobulins, and/or immunosuppressive therapy (including a  $\geq$ 14-day course of systemic corticosteroids) is prohibited during the study.

## **6.8.2.** Permitted During the Study

- If medically necessary (eg, pandemic or outbreak with pandemic potential), licensed influenza or other pandemic vaccines may be given at any time (however, an interval of >14 days prior to or >14 days after study intervention administration is preferred).
- Prescription and nonprescription medications, vitamins, minerals, and herbal remedies are permitted during participation in the study.
- The use of prophylactic antipyretic/pain medication, while permitted, is not recommended on the day of study intervention administration (before or after vaccination). If symptoms develop, the use of antipyretic/pain medication is allowed.
- Inhaled/nebulized, topical (eg, skin, eyes, or ears), or localized injections of corticosteroids (eg, intraarticular or intrabursal administration) are permitted during study participation.

## 6.8.3. Recording Prior and Concomitant Vaccines and Concomitant Treatments

The name and date of administration for all nonstudy vaccinations received from the time of signing of the ICD to Visit 2 will be collected and recorded in the CRF.

Medications taken to treat SAEs from the time of signing of the ICD to Visit 2 will be recorded in the CRF.

# 7. DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 7.1. Discontinuation of Study Intervention

Since this is a single-dose study, this section is not applicable.

## 7.1.1. Participant Discontinuation/Withdrawal From the Study

A participant may withdraw from the study at any time at his/her own request. Reasons for discontinuation from the study include the following:

- Refused further study procedures;
- Lost to follow-up;
- Death;
- Study terminated by sponsor;
- AE;
- Physician decision;
- Pregnancy;
- Protocol deviation;
- Screen failure;
- Withdrawal by participant;
- Medication error without associated AE;
- No longer meets eligibility criteria;
- Other.

If the participant withdraws from the study and also withdraws consent (see Section 7.1.2) for disclosure of future information, no further evaluations should be performed and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

## 7.1.2. Withdrawal of Consent

Participants who request to discontinue receipt of study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him or her or persons previously authorized by the participant to provide this information. Participants should notify the investigator in writing of the decision to withdraw consent from future follow-up, whenever possible. The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is only from further receipt of study intervention or also from study procedures and/or postvaccination study follow-up, and entered on the appropriate CRF page. In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

#### 7.2. Lost to Follow-Up

A participant will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to attend a required study visit:

- The site must attempt to contact the participant and reschedule the missed visit as soon as possible. Counsel the participant on the importance of maintaining the assigned visit schedule, and ascertain whether the participant wishes to and/or should continue in the study;
- Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record;
- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.

#### 8. STUDY ASSESSMENTS AND PROCEDURES

The investigator (or an appropriate delegate at the investigator site) must obtain a signed and dated ICD before performing any study-specific procedures.

The date of birth will be collected to critically evaluate the immune response and safety profile by age.

Study procedures and their timing are summarized in the SoA. Protocol waivers or exemptions are not allowed.

Safety issues should be discussed with the sponsor immediately upon occurrence or awareness to determine whether the participant should continue or discontinue study intervention.

Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.

All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

Every effort should be made to ensure that protocol-required tests and procedures are completed as described. However, it is anticipated that from time to time there may be circumstances outside the control of the investigator that may make it unfeasible to perform the test. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the participant. When a protocol-required test cannot be performed, the investigator will document the reason for the missed test and any corrective and preventive actions that he or she has taken to ensure that required processes are adhered to as soon as possible. The study team must be informed of these incidents in a timely manner.

#### 8.1. Efficacy and/or Immunogenicity Assessments

Not applicable.

#### 8.2. Safety Assessments

A clinical assessment, including medical history and measurement of temperature, will be performed on all participants prior to any vaccination at Visit 1 to determine participant eligibility and to establish a clinical baseline. Significant medical history and significant findings from any physical examination (if performed) will be recorded as medical history in the CRF. Temperature measurement prior to vaccination will be documented and recorded in the CRF.

The participant will be observed for 20 minutes after each study vaccination, and any reactions occurring during that time will be recorded as AEs.

Prompted e-diary events, including local reactions (redness, swelling, and pain at the injection site) at the site of the 13vPnC injection and systemic events (fever, headache, fatigue, muscle pain, and joint pain) that occur 7 days after vaccination (where Day 1 is the

day of vaccination), are graded as described in Section 8.2.3.1 and Section 8.2.3.2. Furthermore, AEs and SAEs will be collected as defined in Section 8.3.

Planned time points for all safety assessments are provided in the SoA. Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety issues.

#### 8.2.1. Physical Examinations

A clinical assessment will be performed at Visit 1. If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, a physical examination will be performed.

Physical examination findings collected during the study will be considered source data and will not be required to be reported, unless otherwise noted. Any untoward physical examination findings that are identified during the active collection period and meet the definition of an AE or SAE (Appendix 3) must be reported according to the processes in Sections 8.3.1 to 8.3.3.

## 8.2.2. Participant Electronic Diary

Participants will be asked to monitor and record local reactions and systemic events using an e-diary (in a provisioned device or an app on a personal device, if available). This allows recording of these assessments only within a fixed time window, thus providing the accurate representation of the participant's experience. Data reported in the e-diary will be transferred electronically to the e-diary vendor, where they will be available for review by investigators, their appropriately qualified designees, and sponsor staff at all times via an internet-based portal. At intervals agreed to by the vendor and Pfizer, these data will be transferred electronically to Pfizer for analysis and reporting.

The daily e-diary data will not be captured in the CRF. However, if a participant is withdrawn because of prompted events reported in the e-diary, the event(s) should be recorded on the AE page of the CRF, regardless of whether the investigator considers the event(s) to be clinically significant.

The investigator or designee must obtain stop dates for any local reactions and specific systemic events that were ongoing on the last day that the e-diary was completed. The stop dates should be entered in the CRF.

Investigators (or an appropriately qualified designee) are required to review the e-diary data online at frequent intervals (daily is optimal) to evaluate participant compliance and reported events as part of the ongoing safety review.

#### 8.2.3. Grading Scale for Prompted Events

The grading scales used in this study to assess prompted events as described below are based on concepts outlined in the FDA CBER guidelines on toxicity grading scales for healthy adult volunteers enrolled in preventive vaccine clinical trials.<sup>31</sup>

#### 8.2.3.1. Local Reactions

For the first 7 days following study vaccination (Days 1 through 7, where Day 1 is the day of vaccination), the participants will be asked to assess redness, swelling, and pain at the injection site and to record the symptoms in the e-diary in the evening. Redness and swelling will be measured in measuring device (caliper) units (range: 1 to 21) and then categorized during analysis as mild, moderate, or severe based on the grading scale in Table 1. Measuring device units can be converted to centimeters according to the following scale: 1 measuring device unit = 0.5 cm. Pain at the vaccine injection site will be assessed by the participant as mild, moderate, or severe according to the grading scale in Table 1. The participant will be prompted to contact the investigator if he/she experiences a severe (Grade 3 or above) local reaction to assess the reaction and perform an unscheduled assessment or visit as appropriate.

Only an investigator is able to classify a participant's local reaction as Grade 4, after physical examination of the participant or documentation from another medically qualified source (eg, emergency room or hospital record). If a participant experiences a Grade 4 local reaction, the investigator must immediately notify the sponsor. Site staff will educate the participants regarding signs and symptoms that would prompt site contact. Grade 4 reactions will be collected as an AE on the CRF. The event will be graded using the AE intensity grading scale (Section 10.3).

The procedure for notification of the sponsor is provided in the ISF or equivalent.

**Table 1. Grading Scales for Local Reactions** 

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 <sup>a</sup> | Grade 4 <sup>b</sup> |
|---|---|---|---|---|
| Redness | 5 to 10 measuring device units = >2.0 to 5.0 cm | 11 to 20 measuring device units = >5.0 to 10.0 cm | >20 measuring device units = >10.0 cm | Necrosis or exfoliative dermatitis |
| Swelling | 5 to 10 measuring<br>device units<br>=<br>>2.0 to 5.0 cm | 11 to 20 measuring device units = >5.0 to 10.0 cm | >20 measuring<br>device units<br>=<br>>10.0 cm | Necrosis |
| Pain at injection site | Does not interfere with activity | Interferes with activity | Prevents daily activity <sup>c</sup> | Emergency room<br>visit or<br>hospitalization for<br>severe injection site<br>pain |

Abbreviation: CRF = case report form.

Note: If the size of the redness and/or swelling falls between 2 measuring device units, the higher measuring device unit number will be recorded in the e-diary.

- a. Participants experiencing Grade 3 local reactions are required to contact the investigator site. In the event that the participant does not call, the investigator will call the participant.
- b. Grade 4 assessment should be made by the investigator; Grade 4 local reactions will not be collected in the e-diary but will be collected as AEs on the CRF, and intensity should be graded using the AE intensity grading scale in Section 10.3.
- c. Prevents daily activity, eg, results in missed days of work or is otherwise incapacitating.

## 8.2.3.2. Systemic Events – Systemic Symptoms and Fever

From Day 1 through Day 7 following vaccination, where Day 1 is the day of vaccination, participants will be asked to assess headache, fatigue, muscle pain, and joint pain and to record the symptoms in the e-diary in the evening. The symptoms will be assessed by the participant as mild, moderate, or severe according to the grading scale in Table 2 below.

Only an investigator is able to classify a participant's systemic event as Grade 4, after physical examination of the participant or documentation from another medically qualified source (eg, emergency room or hospital record) or telephone contact with the participant. If a participant experiences a Grade 4 systemic event, the investigator must immediately notify the sponsor. Grade 4 events will be collected as an AE on the CRF. The event will be graded using the AE intensity grading scale (See Section 10.3).

The procedure for notification of the sponsor is provided in the SRM or equivalent.

**Table 2.** Grading Scales for Systemic Events

| | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 <sup>a</sup> | Grade 4 <sup>b</sup> |
|---|---|---|---|---|
| Fatigue (tiredness) | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room<br>visit or<br>hospitalization for<br>severe fatigue |
| Headache | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room<br>visit or<br>hospitalization for<br>severe headache |
| Muscle pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room<br>visit or<br>hospitalization for<br>severe muscle pain |
| Joint pain | Does not interfere with activity | Some interference with activity | Prevents daily routine activity | Emergency room<br>visit or<br>hospitalization for<br>severe joint pain |

Abbreviation: CRF = case report form.

- a. Prevents daily routine activity, eg, results in missed days of work or is otherwise incapacitating; includes use of narcotics for analgesia.
- b. Grade 4 assessment should be made by the investigator; Grade 4 systemic events will not be collected in the e-diary but will be collected as AEs on the CRF, and intensity should be graded using the AE intensity grading scale in Section 10.3.

#### 8.2.3.2.1. Fever

In order to record information on fever, a digital thermometer will be given to the participant with instructions on how to measure oral temperature at home. Temperature will be collected in the evening daily for 7 days following vaccination (Days 1 through 7, where Day 1 is the day of vaccination) and at any time during the 7 days that fever is suspected. Fever is defined

as an oral temperature of  $\geq 100.4^{\circ}F$  ( $\geq 38.0^{\circ}C$ ). The highest temperature for each day will be recorded in the e-diary. In the event of a fever on Day 7, a temperature will be collected daily until the fever has resolved (1 day of temperature  $< 100.4^{\circ}F$  [ $< 38.0^{\circ}C$ ]) in order to collect a stop date in the CRF. Participants reporting a fever  $> 40.0^{\circ}C$  will be prompted to contact the study site. Study staff may also contact the participant to obtain additional information if a temperature of  $> 102.0^{\circ}F$  ( $> 38.9^{\circ}C$ ) is entered into an e-diary. Temperature will be measured and recorded to 1 decimal place.

Temperatures reported in degrees Fahrenheit will be programmatically converted to degrees Celsius for reporting. Fever will be grouped into ranges for the analysis according to Table 3.

**Table 3.** Ranges for Fever

| ≥38.0°C to 38.4°C |
|----------------------|
| >38.4°C to 38.9°C |
| >38.9°C to 40.0°C |
| >40.0°C <sup>a</sup> |

Note: Fever is defined as a temperature of ≥38.0°C.

a. Participants reporting a fever >40.0°C will be prompted to contact the study site.

## 8.2.4. Clinical Safety Laboratory Assessments

Clinical safety laboratory assessments will not be collected in this study.

#### 8.2.5. Pregnancy Testing

Pregnancy tests may be urine or serum tests, but must have a sensitivity of at least 25 mIU/mL. Pregnancy tests will be performed in WOCBP at the times listed in the SoA, immediately before the administration of each vaccine dose. A negative pregnancy test result will be required prior to the participant's receiving the study intervention. Pregnancy tests may also be repeated if requested by IRBs/ECs or if required by local regulations. In the case of a positive confirmed pregnancy after vaccination, the participant may remain in the study for safety follow-up.

#### 8.3. Adverse Events, Serious Adverse Events, and Other Safety Reporting

The definitions of an AE and an SAE can be found in Appendix 3.

The definitions of device-related safety events (ADEs and SADEs) can be found in Section 10.6. Device deficiencies are covered in Section 8.3.9.

AEs may arise from symptoms or other complaints reported to the investigator by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative), or they may arise from clinical findings of the investigator or other healthcare providers (clinical signs, test results, etc).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible to pursue and obtain adequate information both to determine the outcome and to assess whether the event meets the criteria for classification as an SAE or caused the participant to discontinue the study (see Section 7.1).

During the active collection period as described in Section 8.3.1, each participant will be questioned about the occurrence of AEs in a nonleading manner.

In addition, the investigator may be requested by Pfizer Safety to obtain specific follow-up information in an expedited fashion.

### 8.3.1. Time Period and Frequency for Collecting AE and SAE Information

The time period for actively eliciting and collecting AEs and SAEs ("active collection period") for each participant begins from the time the participant provides informed consent, which is obtained before the participant's participation in the study (ie, before undergoing any study-related procedure and/or receiving study intervention), through and including Visit 2.

Follow-up by the investigator continues throughout and after the active collection period and until the AE or SAE or its sequelae resolve or stabilize at a level acceptable to the investigator.

For participants who are screen failures, the active collection period ends when screen failure status is determined.

If the participant withdraws from the study and also withdraws consent for the collection of future information, the active collection period ends when consent is withdrawn.

If a participant permanently discontinues or temporarily discontinues study because of an AE or SAE, the AE or SAE must be recorded on the CRF and the SAE reported using the Vaccine SAE Reporting Form.

Investigators are not obligated to actively seek information on AEs or SAEs after the participant has concluded study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has completed the study, and he/she considers the event to be reasonably related to the study intervention, the investigator must promptly report the SAE to Pfizer using the Vaccine SAE Reporting Form.

### 8.3.1.1. Reporting SAEs to Pfizer Safety

All SAEs occurring in a participant during the active collection period as described in Section 8.3.1 are reported to Pfizer Safety on the Vaccine SAE Reporting Form immediately upon awareness and under no circumstance should this exceed 24 hours, as indicated in Appendix 3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

## 8.3.1.2. Recording Nonserious AEs and SAEs on the CRF

All nonserious AEs and SAEs occurring in a participant during the active collection period, which begins after obtaining informed consent as described in Section 8.3.1, will be recorded on the AE section of the CRF.

The investigator is to record on the CRF all directly observed and all spontaneously reported AEs and SAEs reported by the participant.

## 8.3.2. Method of Detecting AEs and SAEs

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 3.

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

## 8.3.3. Follow-Up of AEs and SAEs

After the initial AE or SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. For each event, the investigator must pursue and obtain adequate information until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up (as defined in Section 7.2).

In general, follow-up information will include a description of the event in sufficient detail to allow for a complete medical assessment of the case and independent determination of possible causality. Any information relevant to the event, such as concomitant medications and illnesses, must be provided. In the case of a participant death, a summary of available autopsy findings must be submitted as soon as possible to Pfizer Safety.

Further information on follow-up procedures is given in Appendix 3.

#### 8.3.4. Regulatory Reporting Requirements for SAEs

Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities toward the safety of participants and the safety of a study intervention under clinical investigation are met.

The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRBs/ECs, and investigators.

Investigator safety reports must be prepared for SUSARs according to local regulatory requirements and sponsor policy and forwarded to investigators as necessary.

An investigator who receives SUSARs or other specific safety information (eg, summary or listing of SAEs) from the sponsor will review and then file it along with the SRSD(s) for the study and will notify the IRB/EC, if appropriate according to local requirements.

# 8.3.5. Environmental Exposure, Exposure During Pregnancy or Breastfeeding, and Occupational Exposure

Environmental exposure occurs when a person not enrolled in the study as a participant receives unplanned direct contact with or exposure to the study intervention. Such exposure may or may not lead to the occurrence of an AE or SAE. Persons at risk for environmental exposure include healthcare providers, family members, and others who may be exposed. An environmental exposure may include exposure during pregnancy, exposure during breastfeeding, and occupational exposure.

Any such exposure to the study intervention under study is reportable to Pfizer Safety within 24 hours of investigator awareness.

## **8.3.5.1.** Exposure During Pregnancy

An EDP occurs if:

- A female participant is found to be pregnant while receiving or after discontinuing study intervention.
- A male participant who is receiving or has discontinued study intervention exposes a female partner prior to or around the time of conception.
- A female is found to be pregnant while being exposed or having been exposed to study intervention due to environmental exposure. Below are examples of environmental EDP:
  - A female family member or healthcare provider reports that she is pregnant after having been exposed to the study intervention by eg, ingestion, inhalation, or skin contact.

The investigator must report EDP to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The initial information submitted should include the anticipated date of delivery (see below for information related to termination of pregnancy).

• If EDP occurs in a participant or a participant's partner, the investigator must report this information to Pfizer Safety on the Vaccine SAE Reporting Form and an EDP Supplemental Form, regardless of whether an SAE has occurred. Details of the pregnancy will be collected after the start of study intervention and until Visit 2.

• If EDP occurs in the setting of environmental exposure, the investigator must report information to Pfizer Safety using the Vaccine SAE Reporting Form and EDP Supplemental Form. Since the exposure information does not pertain to the participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form is maintained in the investigator site file.

Follow-up is conducted to obtain general information on the pregnancy and its outcome for all EDP reports with an unknown outcome. The investigator will follow the pregnancy until completion (or until pregnancy termination) and notify Pfizer Safety of the outcome as a follow-up to the initial EDP Supplemental Form. In the case of a live birth, the structural integrity of the neonate can be assessed at the time of birth. In the event of a termination, the reason(s) for termination should be specified and, if clinically possible, the structural integrity of the terminated fetus should be assessed by gross visual inspection (unless preprocedure test findings are conclusive for a congenital anomaly and the findings are reported).

Abnormal pregnancy outcomes are considered SAEs. If the outcome of the pregnancy meets the criteria for an SAE (ie, ectopic pregnancy, spontaneous abortion, intrauterine fetal demise, neonatal death, or congenital anomaly in a live-born baby, a terminated fetus, an intrauterine fetal demise, or a neonatal death), the investigator should follow the procedures for reporting SAEs. Additional information about pregnancy outcomes that are reported to Pfizer Safety as SAEs follows:

- Spontaneous abortion including miscarriage and missed abortion;
- Neonatal deaths that occur within 1 month of birth should be reported, without regard to causality, as SAEs. In addition, infant deaths after 1 month should be reported as SAEs when the investigator assesses the infant death as related or possibly related to exposure to the study intervention.

Additional information regarding the EDP may be requested by the sponsor. Further follow-up of birth outcomes will be handled on a case-by-case basis (eg, follow-up on preterm infants to identify developmental delays). In the case of paternal exposure, the investigator will provide the participant with the Pregnant Partner Release of Information Form to deliver to his partner. The investigator must document in the source documents that the participant was given the Pregnant Partner Release of Information Form to provide to his partner.

## 8.3.5.2. Exposure During Breastfeeding

An exposure during breastfeeding occurs if:.

• A female participant is found to be breastfeeding while receiving or after discontinuing study intervention.

• A female is found to be breastfeeding while being exposed or having been exposed to study intervention (ie, environmental exposure). An example of environmental exposure during breastfeeding is a female family member or healthcare provider who reports that she is breastfeeding after having been exposed to the study intervention by eg, ingestion, inhalation, or skin contact.

The investigator must report exposure during breastfeeding to Pfizer Safety within 24 hours of the investigator's awareness, irrespective of whether an SAE has occurred. The information must be reported using the Vaccine SAE Reporting Form. When exposure during breastfeeding occurs in the setting of environmental exposure, the exposure information does not pertain to the participant enrolled in the study, so the information is not recorded on a CRF. However, a copy of the completed Vaccine SAE Reporting Form is maintained in the investigator site file.

An exposure during breastfeeding report is not created when a Pfizer drug specifically approved for use in breastfeeding women (eg, vitamins) is administered in accord with authorized use. However, if the infant experiences an SAE associated with such a drug, the SAE is reported together with the exposure during breastfeeding.

## 8.3.5.3. Occupational Exposure

The investigator must report any instance of occupational exposure to Pfizer Safety within 24 hours of the investigator's awareness using the Vaccine SAE Reporting Form, regardless of whether there is an associated SAE. Since the information about the occupational exposure does not pertain to a participant enrolled in the study, the information is not recorded on a CRF; however, a copy of the completed Vaccine SAE Reporting Form must be maintained in the investigator site file.

#### 8.3.6. Cardiovascular and Death Events

Not applicable.

# 8.3.7. Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs

Not applicable.

#### 8.3.8. Adverse Events of Special Interest

Not applicable.

## 8.3.8.1. Lack of Efficacy

The investigator must report signs, symptoms, and/or clinical sequelae resulting from lack of efficacy.

Lack of efficacy or failure of expected pharmacological action in an approved indication constitutes an SAE and should be reported to Pfizer Safety.

#### 8.3.9. Medical Device Deficiencies

Medical devices being provided for use in this study as the study intervention is supplied in a prefilled syringe. In order to fulfill regulatory reporting obligations worldwide, the investigator is responsible for the detection and documentation of events meeting the definitions of device deficiency that occur during the study with such devices.

The definition of a medical device deficiency can be found in Appendix 6.

Note: AEs and/or SAEs that are associated with a medical device deficiency will follow the same processes as other AEs or SAEs, as outlined in Sections 8.3.1 through 8.3.4 and Appendix 3 of the protocol.

#### 8.3.9.1. Time Period for Detecting Medical Device Deficiencies

Medical device deficiencies that result in an incident will be detected, documented, and reported during all periods of the study in which the medical device is used.

Importantly, reportable device deficiencies are not limited to problems with the device itself but also include incorrect or improper use of the device and even intentional misuse, etc.

If the investigator learns of any device deficiency at any time after a participant has been discharged from the study, and such deficiency is considered reasonably related to a medical device provided for the study, the investigator will promptly notify the sponsor.

The method of documenting medical device deficiencies is provided in Appendix 6.

#### 8.3.9.2. Follow-Up of Medical Device Deficiencies

Follow-up applies to all participants, including those who discontinue study intervention.

The investigator is responsible for ensuring that follow-up includes any supplemental investigations as indicated to elucidate the nature and/or causality of the deficiency.

New or updated information will be recorded on a follow-up form with all changes signed and dated by the investigator.

## 8.3.9.3. Prompt Reporting of Device Deficiencies to the Sponsor

When a device deficiency occurs:

- 1. The investigator notifies the sponsor by telephone or email within 1 business day of determining that the incident meets the protocol definition of a medical device deficiency.
- 2. The device deficiency must be recorded on the Medical Device Complaint form.
- 3. If an AE (either serious or non-serious) associated with the device deficiency occurs, then the AE must be entered into the AE section of the CRF.
4. If an SAE associated with the device deficiency is brought to the attention of the investigator, the investigator must immediately notify Pfizer Safety of the SAE (see Section 8.3.1.1). All relevant details related to the role of the device in the event must be included in the Vaccine SAE Reporting form as outlined in Sections 8.3.1.1 and 8.3.1.2.

The sponsor will be the contact for the receipt of device deficiency information.

#### 8.3.9.4. Regulatory Reporting Requirements for Device Deficiencies

The investigator will promptly report all device deficiencies occurring with any medical device provided for use in the study in order for the sponsor to fulfill the legal responsibility to notify appropriate regulatory authorities and other entities about certain safety information relating to medical devices being used in clinical studies.

The investigator or responsible person according to local requirements (eg, the head of the medical institution), will comply with the applicable local regulatory requirements relating to the reporting of device deficiencies to the IRB/EC.

#### 8.3.10. Medication Errors

Medication errors may result from the administration or consumption of the study intervention by the wrong participant, or at the wrong time, or at the wrong dosage strength, or inadvertent exposure.

Exposures to the study intervention under study may occur in clinical trial settings, such as medication errors.

| Safety Event | Recorded on the CRF | Reported on the Vaccine SAE<br>Reporting Form to Pfizer Safety<br>Within 24 Hours of Awareness |
|---|---|---|
| Medication errors | All (regardless of whether associated with an AE) | Only if associated with an SAE |

#### Medication errors include:

- Medication errors involving participant exposure to the study intervention;
- Potential medication errors or uses outside of what is foreseen in the protocol that do or do not involve the study participant.

Other examples include, but are not limited to:

- The administration of expired study intervention;
- The administration of an incorrect study intervention;
- The administration of an incorrect dosage;
- The administration of study intervention that has undergone temperature excursion from the specified storage range, unless it is determined by the sponsor that the study intervention under question is acceptable for use.

Such medication errors occurring to a study participant are to be captured on the medication error page of the CRF, which is a specific version of the AE page.

In the event of a medication dosing error, the sponsor should be notified within 24 hours.

Whether or not the medication error is accompanied by an AE, as determined by the investigator, the medication error is recorded on the medication error page of the CRF and, if applicable, any associated AE(s), serious and nonserious, are recorded on the AE page of the CRF.

Medication errors should be reported to Pfizer Safety within 24 hours on a Vaccine SAE Reporting Form **only when associated with an SAE.** 

#### **8.4. Pharmacokinetics**

Pharmacokinetic parameters are not evaluated in this study.

#### 8.5. Genetics

#### **8.5.1. Specified Genetics**

Genetics (specified analyses) are not evaluated in this study.

#### 8.6. Biomarkers

Biomarkers are not evaluated in this study.

#### 8.7. Immunogenicity Assessments

Immunogenicity assessments are not included in this study.

#### 8.8. Health Economics

Health economics/medical resource utilization and health economics parameters are not evaluated in this study.

#### 8.9. Study Procedures

The study procedures are summarized in the SoA. The day of Dose 1 is considered to be Day 1. The timing of visit procedures (ie, prior to vaccination and after vaccination) must be maintained; however, there is flexibility in the order in which the procedures can be conducted at each visit. The only exception is that at Visit 1, the ICD must be signed prior to the start of any study procedure.

#### **8.9.1.** Visit 1 (Vaccination 1 – Day 1)

- Obtain a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study before performing any study-specific procedures.
- Assign a participant number via the IRT.
- Obtain and record the participant's demographic information (including date of birth, sex, race, and ethnicity). The complete date of birth (ie, DD-MMM-YYYY) will be collected to critically evaluate the safety profile by age.
- Obtain and record significant medical history, including the presence of chronic conditions (eg, diabetes, asthma, cardiac disease, COPD), and/or medical history of significance, such as relevant surgical procedures.
- Perform a clinical assessment. If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, perform a physical examination and record any findings in the source documents and, if significant, record such findings on the medical history CRF.
- If applicable, instruct the participant to use appropriate contraceptives until 28 days after administration of the study intervention, and document the conversation and the participant's affirmation in the participant's source document.
- Record nonstudy vaccinations as described in Section 6.8.3.
- Measure and record the participant's oral temperature ( ${}^{\circ}F/{}^{\circ}C$ ).
- Ensure and document that all of the inclusion criteria and none of the exclusion criteria are met and that none of the temporary delay criteria are met.
- Prepare 13vPnC according to the IP manual.
- Administer a single 0.5-mL injection of 13vPnC into the deltoid muscle.

- Site staff will observe the participant for 20 minutes after administration of 13vPnC for any reactions. Record any acute reactions (including time of onset) in the participant's source documents, on the AE CRF, and on the Vaccine SAE Reporting Form, as applicable. Record concomitant medications used to treat SAEs.
- Record AEs and SAEs as described in Section 8.3.
- Issue the participant a measuring device to measure 13vPnC injection site reactions and a digital thermometer, and provide instructions on their use.
- Explain the e-diary technologies available for this study (see Section 8.2.2) and assist the participant in downloading the study app, if available, onto the participant's own device or issue a provisioned device if required. Provide instructions on e-diary completion and ask the participant to complete the reactogenicity e-diary each day from Day 1 through Day 7, with Day 1 being the day of vaccination.
- Ask the participant to contact the investigator site staff or investigator as soon as possible during the 7-day postvaccination period if the participant has redness and/or swelling at the 13vPnC injection site measuring >20 measuring device units (>10 cm) or severe injection site pain (prevents daily activity) to determine if the event requires further assessment by the investigator (refer to Section 8.10).
- Ask the participant to contact the investigator site staff or the investigator as soon as possible if they experience any possible Grade 4 prompted local reaction or systemic event within 7 days, after vaccination (refer to Section 8.10).
- Ask the participant to contact the site staff or investigator immediately if any significant illness or medical event (eg, emergency room visit or hospitalization) occurs.
- Provide the participant with the participant contact card containing the study and investigator information.
- Inform the participant that they may be contacted by site staff to obtain additional information on reports of fever >102.0°F (>38.9°C) or Grade 3 events entered into the e-diary.
- Remind the participant to use appropriate contraceptives until 28 days after vaccination, if applicable.
- Schedule an appointment for the participant to return for the next study visit.
- Remind the participant to bring the reactogenicity e-diary to the next visit.
- The investigator or an authorized designee completes the CRF and the source documents and updates the investigational product accountability records.

• The investigator or appropriately qualified designee reviews the e-diary data online at frequent intervals (daily is optimal) for the 7 days (Day 1 is the day of vaccination) following vaccination to evaluate participant compliance and as part of the ongoing safety review.

#### 8.9.2. Visit 2 (Follow-Up – 28 to 42 Days After Vaccination 1 [Study Days 29 to 43])

If a clinic visit is not possible, refer to Section 10.7.1.

- Record nonstudy vaccinations as described in Section 6.8.3.
- Review the participant's e-diary data. Collect stop dates of any e-diary events (local reactions or systemic events) ongoing on the last day that the e-diary was completed and record stop dates in the CRF.
- Collect the e-diary (if applicable) or assist the participant to remove the study application from his or her own personal device, (if applicable).
- If appropriate perform a clinical assessment. If the clinical assessment indicates that a physical examination is necessary to comprehensively evaluate the participant, perform a physical examination and record any findings in the source documents and, if significant, record such findings on the AE CRF.
- Determine if any AEs or SAEs have occurred since the previous visit, follow up on any previously reported events to determine the outcome (ie, record stop dates or confirm if they are still continuing), record as described in Section 8.3, and record concomitant medications used to treat SAEs.
- The investigator or an authorized designee completes the CRF and the source documents.

#### 8.10. Unscheduled Visits

If the participant experiences any possible Grade 4 prompted systemic event or local reaction, fever >104.0°F (>40.0°C), redness or swelling at the injection site measuring >20 measuring device units (>10.0 cm), or severe injection site pain during the 7 days following vaccination, a telephone contact must occur as soon as possible between the investigator or medically qualified designee and the participant to assess if an unscheduled investigator site visit is required. A site visit should be scheduled as soon as possible to assess the extent of the injection site reaction unless any of the following is true:

- The participant is unable to attend the unscheduled visit.
- The reaction is no longer present at the time of the telephone contact.
- The participant recorded an incorrect value in the e-diary (confirmation of an e-diary data entry error).

• The PI or authorized designee determined it was not needed.

This telephone contact will be recorded in the participant's source documentation and the CRF, including the reason the visit was not scheduled, if that was the case.

If the participant is unable to attend the unscheduled visit, or the PI or authorized designee determined it was not needed, any ongoing reactions must be assessed at the next study visit.

During the unscheduled visit, the reactions should be assessed by the investigator or a medically qualified member of the study staff, such as a study physician or a study nurse, as applicable to the investigator's local practice, who will:

- Measure temperature (°F/°C).
- Measure minimum and maximum diameters of redness (if present).
- Measure minimum and maximum diameters of swelling (if present).
- Assess injection site pain (if present) in accordance with the grades provided in Section 8.2.3.1.
- Assess for other findings associated with the reaction and record on the AE page of the CRF, if appropriate.

#### 9. STATISTICAL CONSIDERATIONS

Methodology for summary and statistical analyses of the data collected in this study is described here and further detailed in a SAP, which will be maintained by the sponsor. The SAP may modify what is outlined in the protocol where appropriate; however, any major modifications of the primary endpoint definitions or their analyses will also be reflected in a protocol amendment.

#### 9.1. Statistical Hypotheses

There is no statistical hypothesis planned for this study.

#### 9.1.1. Estimands

The estimand corresponding to the primary safety objective is described in the table in Section 3. In the evaluation of the primary safety objective, missing reactogenicity e-diary data will not be imputed. A partial AE start date (missing day, missing both month and day) will be imputed by assigning the earliest possible start date using all available information, such as the stop date of the AE and the vaccination date(s) from the same participant, following the Pfizer standard of handling an incomplete AE start date. An AE with a completely missing start date is not allowed in the data collection. No other missing information will be imputed in the safety analysis.

#### 9.2. Analysis Sets

For purposes of analysis, the following analysis sets are defined:

| Participant Analysis Set | Description |
|---|---|
| Enrolled in the study | All participants who signed an ICD. |
| Assigned to study intervention | All participants who are assigned an enrollment number in the IWR system. |
| Safety | All participants who receive any study intervention and have safety data assessed after vaccination. |

#### 9.3. Statistical Analyses

The SAP will be developed and finalized before any analyses are performed and will describe the analyses and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary endpoints.

#### 9.3.1. General Considerations

CIs for all endpoints will be presented as 2-sided at the 95% level unless specified otherwise.

All safety analyses will be performed using the safety analysis set for the entire study cohort.

#### 9.3.2. Analysis for Binary Data

Descriptive statistics for categorical variables (eg, proportions) are the percentage (%), the numerator (n) and the denominator (N) used in the percentage calculation, and the 2-sided 95% CIs where applicable.

The exact 95% CI for binary endpoints will be computed using the F distribution (Clopper-Pearson).

#### 9.3.3. Analysis for Continuous Data

Unless otherwise stated, descriptive statistics for continuous variables are n, mean, median, SD, minimum, and maximum.

## 9.3.4. Primary Endpoint(s)/Estimand(s) Analysis

| Objective | Endpoints and Estimands | Statistics |
|---|---|---|
| Safety | <ul> <li>Proportions of participants with local reactions (redness, swelling, and pain at the injection site) within 7 days after vaccination</li> <li>Proportions of participants with systemic events (fever, headache, fatigue, muscle pain, and joint pain) within 7 days after vaccination</li> </ul> | Descriptive summary<br>statistics for participants<br>with each local<br>reaction/systemic event by<br>intensity levels |
| | • Proportions of participants with AEs within 1 month after vaccination | Descriptive summary statistics |
| | • Proportions of participants with SAEs within 1 month after vaccination | Descriptive summary statistics |

## 9.4. Interim Analyses

No formal interim analysis will be conducted for this study.

### 9.5. Sample Size Determination

The sample size of the study is determined primarily based on considerations of accumulating an informative overall safety database. With 200 vaccinated participants, the study will provide a greater than 86% chance of observing at least 1 AE if the true rate is at least 1% (Table 4).

Table 4. Probability of Detecting at Least 1 AE

| Sample Size | True Rate of AEs | Probability of Observing at<br>Least 1 AE |
|-------------|------------------|-------------------------------------------|
| 200 | 0.5% | 63.3% |
| | 1% | 86.6% |
| | 1.5% | 95.1% |

#### 10. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 10.1. Appendix 1: Regulatory, Ethical, and Study Oversight Considerations

#### 10.1.1. Regulatory and Ethical Considerations

This study will be conducted in accordance with the protocol and with the following:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and CIOMS International Ethical Guidelines;
- Applicable ICH GCP guidelines;
- Applicable laws and regulations, including applicable privacy laws.

The protocol, protocol amendments, ICD, SRSD(s), and other relevant documents (eg, advertisements) must be reviewed and approved by the sponsor, submitted to an IRB/EC by the investigator, and reviewed and approved by the IRB/EC before the study is initiated.

Any amendments to the protocol will require IRB/EC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.

Protocols and any substantial amendments to the protocol will require health authority approval prior to initiation except for changes necessary to eliminate an immediate hazard to study participants.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/EC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/EC;
- Notifying the IRB/EC of SAEs or other significant safety findings as required by IRB/EC procedures;
- Providing oversight of the conduct of the study at the site and adherence to requirements of 21 CFR, ICH GCP guidelines, the IRB/EC, European regulation 536/2014 for clinical studies (if applicable), European Medical Device Regulation 2017/745 for clinical device research (if applicable), and all other applicable local regulations.

#### 10.1.1.1. Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

In the event of any prohibition or restriction imposed (ie, clinical hold) by an applicable regulatory authority in any area of the world, or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the study intervention, Pfizer should be informed immediately.

In addition, the investigator will inform Pfizer immediately of any urgent safety measures taken by the investigator to protect the study participants against any immediate hazard, and of any serious breaches of this protocol or of the ICH GCP guidelines that the investigator becomes aware of.

#### 10.1.2. Financial Disclosure

Investigators and subinvestigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### 10.1.3. Informed Consent Process

The investigator or his/her representative will explain the nature of the study, including the risks and benefits, to the participant and answer all questions regarding the study. The participant should be given sufficient time and opportunity to ask questions and to decide whether or not to participate in the trial.

Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, privacy and data protection requirements, where applicable, and the IRB/EC or study center.

The investigator must ensure that each study participant is fully informed about the nature and objective of the study, the sharing of data related to the study, and possible risks associated with participation, including the risks associated with the processing of the participant's personal data.

The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant .

The participant must be informed that his/her medical records may be examined by Clinical Quality Assurance auditors or other authorized personnel appointed by the sponsor, by appropriate IRB/EC members, and by inspectors from regulatory authorities.

The investigator further must ensure that each study participant is fully informed about his or her right to access and correct his or her personal data and to withdraw consent for the processing of his or her personal data.

The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date on which the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICD.

Participants must be reconsented to the most current version of the ICD(s) during their participation in the study.

A copy of the ICD(s) must be provided to the participant.

#### 10.1.4. Data Protection

All parties will comply with all applicable laws, including laws regarding the implementation of organizational and technical measures to ensure protection of participant data.

Participants' personal data will be stored at the study site in encrypted electronic and/or paper form and will be password-protected or secured in a locked room to ensure that only authorized study staff have access. The study site will implement appropriate technical and organizational measures to ensure that the personal data can be recovered in the event of disaster. In the event of a potential personal data breach, the study site will be responsible for determining whether a personal data breach has in fact occurred and, if so, providing breach notifications as required by law.

To protect the rights and freedoms of participants with regard to the processing of personal data, participants will be assigned a single, participant-specific numerical code. Any participant records or data sets that are transferred to the sponsor will contain the numerical code; participant names will not be transferred. All other identifiable data transferred to the sponsor will be identified by this single, participant-specific code. The study site will maintain a confidential list of participants who participated in the study, linking each participant's numerical code to his or her actual identity and medical record ID. In case of data transfer, the sponsor will protect the confidentiality of participants' personal data consistent with the clinical study agreement and applicable privacy laws.

#### 10.1.5. Committees Structure



#### 10.1.6. Dissemination of Clinical Study Data

Pfizer fulfills its commitment to publicly disclose clinical study results through posting the results of studies on www.clinicaltrials.gov (ClinicalTrials.gov), the EudraCT, and/or www.pfizer.com, and other public registries in accordance with applicable local laws/regulations. In addition, Pfizer reports study results outside of the requirements of local laws/regulations pursuant to its SOPs.

In all cases, study results are reported by Pfizer in an objective, accurate, balanced, and complete manner and are reported regardless of the outcome of the study or the country in which the study was conducted.

#### www.clinicaltrials.gov

Pfizer posts clinical trial results on www.clinicaltrials.gov for Pfizer-sponsored interventional studies (conducted in patients) that evaluate the safety and/or efficacy of a product, regardless of the geographical location in which the study is conducted. These results are submitted for posting in accordance with the format and timelines set forth by US law.

#### EudraCT

Pfizer posts clinical trial results on EudraCT for Pfizer-sponsored interventional studies in accordance with the format and timelines set forth by EU requirements.

#### www.pfizer.com

Pfizer posts public disclosure synopses (CSR synopses in which any data that could be used to identify individual participants have been removed) on www.pfizer.com for Pfizer-sponsored interventional studies at the same time the corresponding study results are posted to www.clinicaltrials.gov.

#### Documents within marketing authorization packages/submissions

Pfizer complies with the European Union Policy 0070, the proactive publication of clinical data to the EMA website. Clinical data, under Phase 1 of this policy, includes clinical overviews, clinical summaries, CSRs, and appendices containing the protocol and protocol amendments, sample CRFs, and statistical methods. Clinical data, under Phase 2 of this policy, includes the publishing of individual participant data. Policy 0070 applies to new marketing authorization applications submitted via the centralized procedure since 01 January 2015 and applications for line extensions and for new indications submitted via the centralized procedure since 01 July 2015.

#### Data sharing

Pfizer provides researchers secure access to patient-level data or full CSRs for the purposes of "bona-fide scientific research" that contributes to the scientific understanding of the disease, target, or compound class. Pfizer will make data from these trials available 24 months after study completion. Patient-level data will be anonymized in accordance with applicable privacy laws and regulations. CSRs will have personally identifiable information redacted.

Data requests are considered from qualified researchers with the appropriate competencies to perform the proposed analyses. Research teams must include a biostatistician. Data will not be provided to applicants with significant conflicts of interest, including individuals requesting access for commercial/competitive or legal purposes.

#### 10.1.7. Data Quality Assurance

All participant data relating to the study will be recorded on printed or electronic CRF unless transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

Guidance on completion of CRFs will be provided in the CRF Completion Requirements document.

The investigator must ensure that the CRFs are securely stored at the study site in encrypted electronic form and are password to prevent access by unauthorized third parties.

QTLs are predefined parameters that are monitored during the study. Important deviations from the QTLs and any remedial actions taken will be summarized in the clinical study report.

The investigator must permit study-related monitoring, audits, IRB/EC review, and regulatory agency inspections and provide direct access to source data documents. This verification may also occur after study completion. It is important that the investigator(s) and their relevant personnel are available during the monitoring visits and possible audits or inspections and that sufficient time is devoted to the process.

Monitoring details describing strategy, including definition of study critical data items and processes (eg, risk-based initiatives in operations and quality such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, virtual, or on-site monitoring), are provided in the data management plan maintained and utilized by the sponsor or designee.

The sponsor or designee is responsible for the data management of this study, including quality checking of the data.

Records and documents, including signed ICDs, pertaining to the conduct of this study must be retained by the investigator for 15 years after study completion unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor. The investigator must ensure that the records continue to be stored securely for as long as they are maintained.

When participant data are to be deleted, the investigator will ensure that all copies of such data are promptly and irrevocably deleted from all systems.

The investigator(s) will notify the sponsor or its agents immediately of any regulatory retain notification in relation to the study. Furthermore, the investigator will cooperate with the sponsor or its agents to prepare the investigator site for the inspection and will allow the sponsor or its agent, whenever feasible, to be present during the inspection. The investigator site and investigator will promptly resolve any discrepancies that are identified between the study data and the participant's medical records. The investigator will promptly provide copies of the inspection findings to the sponsor or its agent. Before response submission to the regulatory authorities, the investigator will provide the sponsor or its agents with an opportunity to review and comment on responses to any such findings.

#### 10.1.8. Source Documents

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator site.

Data reported on the CRF or entered in the eCRF that are from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.

Definition of what constitutes source data and its origin can be found in the clinical monitoring plan, which is maintained by the sponsor.

Description of the use of the computerized system is documented in the data management plan, which is maintained by the sponsor.

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.

Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorized site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP guidelines, and all applicable regulatory requirements.

#### 10.1.9. Study and Site Start and Closure

The study start date is the date on which the clinical study will be open for recruitment of participants.

The first act of recruitment is the date of the first participant's first visit and will be the study start date.

The sponsor designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time upon notification to the sponsor or designee if requested to do so by the responsible IRB/EC or if such termination is required to protect the health of study participants.

Reasons for the early closure of a study site by the sponsor may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/EC or local health authorities, the sponsor's procedures, or the ICH GCP guidelines;
- Inadequate recruitment of participants by the investigator;
- Discontinuation of further study intervention development.

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the ECs/IRBs, the regulatory authorities, and any CRO(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

Study termination is also provided for in the clinical study agreement. If there is any conflict between the contract and this protocol, the contract will control as to termination rights.

#### 10.1.10. Publication Policy

The results of this study may be published or presented at scientific meetings by the investigator after publication of the overall study results or 1 year after the end of the study (or study termination), whichever comes first.

The investigator agrees to refer to the primary publication in any subsequent publications, such as secondary manuscripts, and submits all manuscripts or abstracts to the sponsor 30 days before submission. This allows the sponsor to protect proprietary information and to provide comments, and the investigator will, on request, remove any previously undisclosed confidential information before disclosure, except for any study- or Pfizer intervention—related information necessary for the appropriate scientific presentation or understanding of the study results.

For all publications relating to the study, the investigator will comply with recognized ethical standards concerning publications and authorship, including those established by the International Committee of Medical Journal Editors.

The sponsor will comply with the requirements for publication of the overall study results covering all investigator sites. In accordance with standard editorial and ethical practice, the sponsor will support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.

Authorship of publications for the overall study results will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

If publication is addressed in the clinical study agreement, the publication policy set out in this section will not apply.

#### 10.1.11. Sponsor's Qualified Medical Personnel

The contact information for the sponsor's appropriately qualified medical personnel for the study is documented in the study contact list located in the supporting study documentation/study portal or other electronic system.

To facilitate access to appropriately qualified medical personnel for study-related medical questions or problems, participants are provided with an Emergency Contact Card (ECC) at the time of informed consent. The ECC contains, at a minimum, (a) protocol and study intervention identifiers, (b) participant's study identification number, (c) site emergency phone number active 24 hours/day, 7 days per week, and (d) Pfizer Call Center number.

The ECC is intended to augment, not replace, the established communication pathways between the investigator, site staff, and study team. The ECC is to be used by healthcare professionals not involved in the research study only, as a means of reaching the investigator or site staff related to the care of a participant. The Pfizer Call Center number should only be used when the investigator and site staff cannot be reached. The Pfizer Call Center number is not intended for use by the participant directly; if a participant calls that number directly, he or she will be directed back to the investigator site.

## 10.2. Appendix 2: Clinical Laboratory Tests

Not applicable.

# 10.3. Appendix 3: Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting

#### 10.3.1. Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
- Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

#### **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or other safety assessments (eg, ECG, radiological scans, vital sign measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgment of the investigator. Any abnormal laboratory test results that meet any of the conditions below must be recorded as an AE:
  - Is associated with accompanying symptoms.
  - Requires additional diagnostic testing or medical/surgical intervention.
  - Leads to a change in study dosing (outside of any protocol-specified dose adjustments) or discontinuation from the study, significant additional concomitant drug treatment, or other therapy.
- Exacerbation of a chronic or intermittent preexisting condition, including either an increase in frequency and/or intensity of the condition.
- New condition detected or diagnosed after study intervention administration, even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE or SAE unless it is an intentional overdose taken with possible

suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

#### **Events NOT Meeting the AE Definition**

- Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (eg, endoscopy, appendectomy): the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2. Definition of an SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed below:

#### a. Results in death

#### b. Is life-threatening

The term "life-threatening" in the definition of "serious" refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it were more severe.

#### c. Requires inpatient hospitalization or prolongation of existing hospitalization

In general, hospitalization signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is

serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a preexisting condition that did not worsen from baseline is not considered an AE.

#### d. Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance, such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (eg, sprained ankle), that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

# f. Is a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic, is considered serious.

The event may be suspected from clinical symptoms or laboratory findings indicating an infection in a participant exposed to a Pfizer product. The terms "suspected transmission" and "transmission" are considered synonymous. These cases are considered unexpected and handled as serious expedited cases by pharmacovigilance personnel. Such cases are also considered for reporting as product defects, if appropriate.

#### g. Other situations:

- Medical or scientific judgment should be exercised by the investigator in deciding
  whether SAE reporting is appropriate in other situations, such as significant
  medical events that may jeopardize the participant or may require medical or
  surgical intervention to prevent one of the other outcomes listed in the above
  definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

# 10.3.3. Recording/Reporting and Follow-Up of AEs and/or SAEs During the Active Collection Period

#### AE and SAE Recording/Reporting

The table below summarizes the requirements for recording AEs on the CRF and for reporting SAEs on the Vaccine SAE Reporting Form to Pfizer Safety throughout the active collection period. These requirements are delineated for 3 types of events: (1) SAEs; (2) nonserious AEs; and (3) exposure to the study intervention under study during pregnancy or breastfeeding, and occupational exposure.

It should be noted that the Vaccine SAE Reporting Form for reporting of SAE information is not the same as the AE page of the CRF. When the same data are collected, the forms must be completed in a consistent manner. AEs should be recorded using concise medical terminology and the same AE term should be used on both the CRF and the Vaccine SAE Reporting Form for reporting of SAE information.

| Safety Event | Recorded on the CRF | Reported on the Vaccine<br>SAE Reporting Form to<br>Pfizer Safety Within 24<br>Hours of Awareness |
|---|---|---|
| SAE | All | All |
| Nonserious AE | All | None |
| Exposure to the study intervention under study during pregnancy or breastfeeding. | All AEs or SAEs associated with exposure during pregnancy or breastfeeding. | All instances of EDP are reported (whether or not there is an associated SAE).* |
| | Note: Instances of EDP or EDB not associated with an AE or SAE are not captured in the CRF. | All instances of EDB are reported (whether or not there is an associated SAE).** |
| Environmental or occupational exposure to the product under study to a non-participant (not involving EDP or EDB). | None. Exposure to a study non-participant is not collected on the CRF. | The exposure (whether or not there is an associated AE or SAE) must be reported.*** |

<sup>\*</sup> EDP (with or without an associated AE or SAE): any pregnancy information is reported to Pfizer Safety using the Vaccine SAE Reporting Form and EDP Supplemental Form; if the EDP is associated with an SAE, then the SAE is reported to Pfizer Safety using the Vaccine SAE Reporting Form.

<sup>\*\*</sup> **EDB** is reported to Pfizer Safety using the Vaccine SAE Reporting Form, which would also include details of any SAE that might be associated with the EDB.

- \*\*\* Environmental or occupational exposure: AEs or SAEs associated with occupational exposure are reported to Pfizer Safety using the Vaccine SAE Reporting Form.
  - When an AE or SAE occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.
  - The investigator will then record all relevant AE or SAE information in the CRF.
  - It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of completion of the Vaccine SAE Reporting Form/AE or SAE CRF page.
  - There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.
  - The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE or SAE.

#### **Assessment of Intensity**

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to 1 of the following categories: .

| GRADE | If required on the AE page of the CRF, the investigator will use the adjectives MILD, MODERATE, SEVERE, or LIFE-THREATENING to describe the maximum intensity of the AE. For purposes of consistency, these intensity grades are defined as follows: | |
|---|---|---|
| 1 | MILD | Does not interfere with participant's usual function. |
| 2 | MODERATE | Interferes to some extent with participant's usual function. |
| 3 | SEVERE | Interferes significantly with participant's usual function. |
| 4 | LIFE-THREATENING | Life-threatening consequences; urgent intervention indicated. |

#### **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE or SAE. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration, will be considered and investigated.
- The investigator will also consult the IB and/or product information, for marketed products, in his/her assessment.
- For each AE or SAE, the investigator <u>must</u> document in the medical notes that he/she has reviewed the AE or SAE and has provided an assessment of causality.

- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.
- If the investigator does not know whether or not the study intervention caused the event, then the event will be handled as "related to study intervention" for reporting purposes, as defined by the sponsor. In addition, if the investigator determines that an SAE is associated with study procedures, the investigator must record this causal relationship in the source documents and CRF, and report such an assessment in the dedicated section of the Vaccine SAE Reporting Form and in accordance with the SAE reporting requirements.

#### Follow-Up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations, as medically indicated or as requested by the sponsor, to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- If a participant dies during participation in the study or during a recognized follow-up period, the investigator will provide Pfizer Safety with a copy of any postmortem findings, including histopathology.
- New or updated information will be recorded in the originally submitted documents.
- The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 10.3.4. Reporting of SAEs

#### SAE Reporting to Pfizer Safety via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to Pfizer Safety will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) to report the event within 24 hours.
- The site will enter the SAE data into the electronic system as soon as the data become available.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section) or to Pfizer Safety by telephone.

#### SAE Reporting to Pfizer Safety via Vaccine SAE Reporting Form

- Facsimile transmission of the Vaccine SAE Reporting Form is the preferred method to transmit this information to Pfizer Safety.
- In circumstances when the facsimile is not working, notification by telephone is acceptable with a copy of the Vaccine SAE Reporting Form sent by overnight mail or courier service.
- Initial notification via telephone does not replace the need for the investigator to complete and sign the Vaccine SAE Reporting Form pages within the designated reporting time frames.

#### 10.4. Appendix 4: Contraceptive and Barrier Guidance

#### 10.4.1. Male Participant Reproductive Inclusion Criteria

Male participants are eligible to participate if they agree to the following requirements during the intervention period and for at least 28 days after the last dose of study intervention:

• Refrain from donating sperm.

#### PLUS either:

 Be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

OR

- Must agree to use contraception/barrier as detailed below:
  - Agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
- In addition to male condom use, a highly effective method of contraception may be considered in WOCBP partners of male participants (refer to the list of highly effective methods below in Section 10.4.4).

#### 10.4.2. Female Participant Reproductive Inclusion Criteria

A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:

• Is not a WOCBP (see definitions below in Section 10.4.3).

OR

• Is a WOCBP and using an <u>acceptable</u> contraceptive method as described below during the intervention period (for a minimum of 28 days after the last dose of study intervention). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

#### 10.4.3. Woman of Childbearing Potential

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile (see below).

If fertility is unclear (eg, amenorrhea in adolescents or athletes) and a menstrual cycle cannot be confirmed before the first dose of study intervention, additional evaluation should be considered.

Women in the following categories are not considered WOCBP:

- 1. Premenarchal.
- 2. Premenopausal female with 1 of the following:
  - Documented hysterectomy;
  - Documented bilateral salpingectomy;
  - Documented bilateral oophorectomy.

For individuals with permanent infertility due to an alternate medical cause other than the above, (eg, mullerian agenesis, androgen insensitivity), investigator discretion should be applied to determining study entry.

Note: Documentation for any of the above categories can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview. The method of documentation should be recorded in the participant's medical record for the study.

#### 3. Postmenopausal female:

- A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. In addition:
  - A high FSH level in the postmenopausal range must be used to confirm a postmenopausal state in women under 60 years of age and not using hormonal contraception or HRT.
  - A female on HRT and whose menopausal status is in doubt will be required to use one of the nonestrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

#### 10.4.4. Contraception Methods

Contraceptive use by men or women should be consistent with local availability/regulations regarding the use of contraceptive methods for those participating in clinical trials.

- 1. Implantable progestogen-only hormone contraception associated with inhibition of ovulation.
- 2. Intrauterine device.
- 3. Intrauterine hormone-releasing system.
- 4. Bilateral tubal occlusion (eg, bilateral tubal ligation).
- 5. Vasectomized partner:
  - A vasectomized partner is a highly effective contraceptive method provided that the partner is the sole sexual partner of the woman of childbearing potential and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used. The spermatogenesis cycle is approximately 90 days.
- 6. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:
  - Oral;
  - Intravaginal;
  - Transdermal.
- 7. Progestogen-only hormone contraception associated with inhibition of ovulation:
  - Oral;
  - Injectable.
- 8. Sexual abstinence:
  - Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study intervention. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
- 9. Progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action.

- 10. Male or female condom with or without spermicide.
- 11. Cervical cap, diaphragm, or sponge with spermicide.
- 12. A combination of male condom with either cervical cap, diaphragm, or sponge with spermicide (double-barrier methods).

# 10.5. Appendix 5: Liver Safety: Suggested Actions and Follow-Up Assessments Potential Cases of Drug-Induced Liver Injury

Humans exposed to a drug who show no sign of liver injury (as determined by elevations in transaminases) are termed "tolerators," while those who show transient liver injury but adapt are termed "adaptors." In some participants, transaminase elevations are a harbinger of a more serious potential outcome. These participants fail to adapt and therefore are "susceptible" to progressive and serious liver injury, commonly referred to as DILI. Participants who experience a transaminase elevation above 3 × ULN should be monitored more frequently to determine if they are "adaptors" or are "susceptible."

LFTs are not required as a routine safety monitoring procedure in this study. However, should an investigator deem it necessary to assess LFTs because a participant presents with clinical signs/symptoms, such LFT results should be managed and followed as described below.

In the majority of DILI cases, elevations in AST and/or ALT precede TBili elevations (>2 × ULN) by several days or weeks. The increase in TBili typically occurs while AST/ALT is/are still elevated above 3 × ULN (ie, AST/ALT and TBili values will be elevated within the same laboratory sample). In rare instances, by the time TBili elevations are detected, AST/ALT values might have decreased. This occurrence is still regarded as a potential DILI. Therefore, abnormal elevations in either AST OR ALT in addition to TBili that meet the criteria outlined below are considered potential DILI (assessed per Hy's law criteria) cases and should always be considered important medical events, even before all other possible causes of liver injury have been excluded.

The threshold of laboratory abnormalities for a potential DILI case depends on the participant's individual baseline values and underlying conditions. Participants who present with the following laboratory abnormalities should be evaluated further as potential DILI (Hy's law) cases to definitively determine the etiology of the abnormal laboratory values:

- Participants with AST/ALT and TBili baseline values within the normal range who subsequently present with AST OR ALT values >3 × ULN AND a TBili value >2 × ULN with no evidence of hemolysis and an alkaline phosphatase value <2 × ULN or not available.</li>
- For participants with baseline AST **OR** ALT **OR** TBili values above the ULN, the following threshold values are used in the definition mentioned above, as needed, depending on which values are above the ULN at baseline:
  - Preexisting AST or ALT baseline values above the normal range: AST or ALT values >2 times the baseline values AND >3 × ULN; or >8 × ULN (whichever is smaller).

• Preexisting values of TBili above the normal range: TBili level increased from baseline value by an amount of at least 1 × ULN **or** if the value reaches >3 × ULN (whichever is smaller).

Rises in AST/ALT and TBili separated by more than a few weeks should be assessed individually based on clinical judgment; any case where uncertainty remains as to whether it represents a potential Hy's law case should be reviewed with the sponsor.

The participant should return to the investigator site and be evaluated as soon as possible, preferably within 48 hours from awareness of the abnormal results. This evaluation should include laboratory tests, detailed history, and physical assessment.

In addition to repeating measurements of AST and ALT and TBili for suspected Hy's law cases, additional laboratory tests should include albumin, CK, direct and indirect bilirubin, GGT, PT/INR, total bile acids, and alkaline phosphatase. Consideration should also be given to drawing a separate tube of clotted blood and an anticoagulated tube of blood for further testing, as needed, for further contemporaneous analyses at the time of the recognized initial abnormalities to determine etiology. A detailed history, including relevant information, such as review of ethanol, acetaminophen/paracetamol (either by itself or as a coformulated product in prescription or over-the-counter medications), recreational drug, or supplement (herbal) use and consumption, family history, sexual history, travel history, history of contact with a jaundiced person, surgery, blood transfusion, history of liver or allergic disease, and potential occupational exposure to chemicals, should be collected. Further testing for acute hepatitis A, B, C, D, and E infection, liver imaging (eg, biliary tract), and collection of serum samples for acetaminophen/paracetamol drug and/or protein adduct levels may be warranted.

All cases demonstrated on repeat testing as meeting the laboratory criteria of AST/ALT and TBili elevation defined above should be considered potential DILI (Hy's law) cases if no other reason for the LFT abnormalities has yet been found. Such potential DILI (Hy's law) cases are to be reported as SAEs, irrespective of availability of all the results of the investigations performed to determine etiology of the LFT abnormalities.

A potential DILI (Hy's law) case becomes a confirmed case only after all results of reasonable investigations have been received and have excluded an alternative etiology.

# 10.6. Appendix 6: AEs, ADEs, SAEs, SADEs, USADEs, and Device Deficiencies: Definitions and Procedures for Recording, Evaluating, Follow-Up, and Reporting in Medical Device Studies

#### **Definitions of a Medical Device Deficiency**

The definitions and procedures detailed in this appendix are in accordance with ISO 14155 and the EU MDR 2017/745 for clinical device research (if applicable).

Both the investigator and the sponsor will comply with all local reporting requirements for medical devices.

The detection and documentation procedures described in this protocol apply to all sponsor medical devices provided for use in the study (see Section 6.1.2 for the list of sponsor medical devices).

#### 10.6.1. Definition of AE and ADE

#### AE and ADE Definition

- An AE is defined in Appendix 3 (Section 10.3.1).
- An ADE is defined as an AE related to the use of an investigational medical device.
   This definition includes any AEs resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device as well as any event resulting from use error or from intentional misuse of the investigational medical device.

#### 10.6.2. Definition of SAE, SADE, and USADE

#### **SAE Definition**

• An SAE is defined in Appendix 3 (Section 10.3.2).

#### **SADE Definition**

- An SADE is defined as an adverse device effect that has resulted in any of the consequences characteristic of an SAE.
- Any device deficiency that might have led to an SAE if appropriate action had not been taken, intervention had not occurred, or circumstances had been less fortunate.

#### **USADE Definition**

• A USADE is a serious adverse device effect that by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis management file.

#### **10.6.3.** Definition of Device Deficiency

#### **Device Deficiency Definition**

• A device deficiency is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. Device deficiencies include malfunctions, use errors, and inadequate information supplied by the manufacturer.

#### 10.6.4. Recording/Reporting and Follow-Up of Medical Device Deficiencies

#### **Device Deficiency Recording**

- When a device deficiency occurs, it is the responsibility of the investigator to review all documentation (eg, hospital progress notes, laboratory reports, and diagnostic reports) related to the event.
- The investigator will then record all relevant device deficiency information in the participant's medical records, in accordance with the investigator's normal clinical practice and will also capture the required information on the Medical Device Complaint form.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to Pfizer Safety in lieu of following the reporting process described in the Medical Device Complaint form.
- There may be instances when copies of medical records for certain cases are requested by Pfizer Safety. In this case, all participant identifiers, with the exception of the participant number, will be redacted on the copies of the medical records before submission to Pfizer Safety.
- If the investigator determines that the medical device deficiency may have injured the participant (ie, the medical device deficiency is associated with an AE or SAE), then the investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis will be documented in the participant's medical record and recorded as the AE or SAE rather than the individual signs/symptoms. Requirements for

recording and reporting an AE or SAE are provided in Appendix 3 (Section 10.3.3).

- For device deficiencies, it is very important that the investigator describes any corrective or remedial actions taken to prevent recurrence of the incident.
  - A remedial action is any action other than routine maintenance or servicing of a
    medical device where such action is necessary to prevent recurrence of a device
    deficiency. This includes any amendment to the device design to prevent
    recurrence.

#### Assessment of Causality Occurring in Conjunction With a Medical Device Deficiency

- If an AE or SAE has occurred in conjunction with a medical device deficiency, the investigator must assess the relationship between each occurrence of the AE or SAE and the medical device deficiency. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.
- The investigator will also consult the local package insert in his/her assessment.
- For each device deficiency, the investigator <u>must</u> document in the medical notes that he/she has reviewed the device deficiency and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

#### Follow-Up of Medical Device Deficiency

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations, as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the device deficiency as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other healthcare providers.
- New or updated information regarding the nature of the device deficiency will be recorded in the originally completed Medical Device Complaint form.
- New or updated information regarding any SAE that was potentially associated with the medical device deficiency will be submitted to Pfizer Safety on the Vaccine SAE Reporting Form within 24 hours of receipt of the information, according to the requirements provided in Appendix 3.

#### 10.6.5. Reporting of SAEs

Reporting of an SAE to Pfizer Safety must be performed according to the processes described in Appendix 3 (Section 10.3.4).

#### 10.6.6. Reporting of SADEs

#### **SADE Reporting to Pfizer Safety**

Note: There are additional reporting obligations for medical device deficiencies that are potentially related to SAEs (ie, a SADE) that must fulfill the legal responsibility to notify appropriate regulatory authorities and other entities about certain safety information relating to medical devices being used in clinical studies.

- Any device deficiency that is associated with an SAE must be reported to the sponsor within 24 hours after the investigator determines that the event meets the definition of a device deficiency.
- The sponsor shall review all device deficiencies and determine and document in writing whether they could have led to an SAE. These shall be reported to the regulatory authorities and IRBs/ECs as required by national regulations.

#### 10.7. Appendix 7: Alternative Measures During Public Emergencies

The alternative study measures described in this section are to be followed during public emergencies, including the COVID-19 pandemic. This appendix applies for the duration of the COVID-19 pandemic and will become effective for other public emergencies only upon written notification from Pfizer.

Use of these alternative study measures is expected to cease upon the return of business as usual (including the lifting of any quarantines and travel bans/advisories).

#### 10.7.1. Telehealth Visits

In the event that in-clinic study visits cannot be conducted, every effort should be made to follow up on the safety of study participants at scheduled visits per the Schedule of Activities or unscheduled visits. Telehealth visits may be used to continue to assess participant safety and collect data points. Telehealth includes the exchange of healthcare information and services via telecommunication technologies (eg, audio, video, video-conferencing software) remotely, allowing the participant and the investigator to communicate on aspects of clinical care, including medical advice, reminders, education, and safety monitoring. The following assessments must be performed during a telehealth visit:

- Review and record any AEs and SAEs since the last contact. Refer to Section 8.3.
- Review any new concomitant medications or changes in concomitant medications since the last contact. Record details of medication to treat any SAE.
- Review and record contraceptive method and results of pregnancy testing. Confirm that the participant is adhering to the contraception method(s) required in the protocol. Refer to Section 10.4 of this appendix regarding pregnancy tests.

Study participants must be reminded to promptly notify site staff about any change in their health status.

## 10.8. Appendix 8: Abbreviations

The following is a list of abbreviations that may be used in the protocol.

| Abbreviation | Term |
|---|---|
| 13vPnC | 13-valent pneumococcal conjugate vaccine |
| ACIP | Advisory Committee on Immunization Practices |
| ADE | adverse device effect |
| AE | adverse event |
| ALT | alanine aminotransferase |
| AOM | acute otitis media |
| арр | application |
| ALT | alanine aminotransferase |
| AST | aspartate aminotransferase |
| CAP | community-acquired pneumonia |
| CAPiTA | Community-Acquired Pneumonia Immunization Trial in Adults |
| CBER | Center for Biologics Evaluation and Research |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CIOMS | Council for International Organizations of Medical Sciences |
| CK | creatine kinase |
| CONSORT | Consolidated Standards of Reporting Trials |
| COPD | chronic obstructive pulmonary disease |
| COVID-19 | coronavirus disease 2019 |
| CRF | case report form |
| CRM <sub>197</sub> | cross-reactive material 197 |
| CRO | contract research organization |
| CSF | cerebrospinal fluid |
| CSR | clinical study report |
| DCGI | Drug Controller General of India |
| DILI | drug-induced liver injury |
| CCI | |
| EC | ethics committee |
| ECC | emergency contact card |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| e-diary | electronic diary |
| EDB | exposure during breastfeeding |
| EDP | exposure during pregnancy |
| EMA | European Medicines Agency |
| EU | European Union |
| EU MDR | European Union Medical Device Regulation |
| EudraCT | European Clinical Trials Database |
| FDA | Food and Drug Administration |

| Abbreviation | Term |
|--------------|-------------------------------------------------|
| FSH | follicle-stimulating hormone |
| GCP | Good Clinical Practice |
| GGT | gamma-glutamyl transferase |
| HRT | hormone replacement therapy |
| IB | investigator's brochure |
| ICD | informed consent document |
| ICH | International Council for Harmonisation |
| ID | identification |
| IND | investigational new drug application |
| INR | international normalized ratio |
| IP manual | investigational product manual |
| IPAL | Investigational Product Accountability Log |
| IPD | invasive pneumococcal disease |
| IRB | institutional review board |
| IRT | interactive response technology |
| ISO | International Organization for Standardization |
| ISF | investigator site file |
| IWR | interactive Web-based response |
| LFT | liver function test |
| N/A | not applicable |
| PASS | postauthorization safety study |
| PPSV23 | 23-valent pneumococcal polysaccharide vaccine |
| PT | prothrombin time |
| QTL | quality tolerance limit |
| SADE | serious adverse device effect |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SARS-CoV-2 | severe acute respiratory syndrome coronavirus 2 |
| SD | standard deviation |
| SEC | subject expert committee |
| SoA | schedule of activities |
| SOP | standard operating procedure |
| SRSD | single reference safety document |
| SUSAR | suspected unexpected serious adverse reaction |
| TBili | total bilirubin |
| ULN | upper limit of normal |
| US | United States |
| USADE | unanticipated serious adverse device effect |
| VT | vaccine-type |
| WOCBP | woman/women of childbearing potential |

#### 11. REFERENCES

- Iyer AS, Ohtola JA, Westerink MAJ. Age-related immune response to pneumococcal polysaccharide vaccination: lessons for the clinic. Expert Rev Vaccines. 2015;14(1):85-97.
- Nuorti JP, Butler JC, Farley MM, et al. Cigarette smoking and invasive pneumococcal disease. N Engl J Med. 2000;342(10):681-9.
- Malik A, Taneja D. Conjugate pneumococcal vaccines: need and choice in India. Indian J Community Med. 2013;38(4):189-91.
- Gierke R, Wodi P, Kobayashi M. Pneumococcal disease. Chapter 17. In: Hall E, Wodi AP, Hamborsky J, et al, eds. Epidemiology and prevention of vaccine-preventable diseases. 14th ed. Washington, DC: Public Health Foundation; 2021;255-74. Available from: https://www.cdc.gov/vaccines/pubs/pinkbook/downloads/pneumo.pdf. Accessed: 23 Sep 2021.
- Thomas K, Mukkai Kesavan L, Veeraraghavan B, et al. Invasive pneumococcal disease associated with high case fatality in India. J Clin Epidemiol. 2013;66(1):36-43.
- Jayaraman R, Varghese R, Kumar JL, et al. Invasive pneumococcal disease in Indian adults: 11 years' experience. J Microbiol Immunol Infect. 2019;52(5):736-42.
- Dey AB, Nagarkar KM, Kumar V. Clinical presentation and predictors of outcome in adult patients with community-acquired pneumonia. Natl Med J India. 1997;10(4):169-72.
- Bansal S, Kashyap S, Pal LS, et al. Clinical and bacteriological profile of community acquired pneumonia in Shimla, Himachal Pradesh. Indian J Chest Dis Allied Sci. 2004;46(1):17-22.
- Oberoi A, Aggarwal A. Bacteriological profile, serology and antibiotic sensitivity pattern of micro-organisms from community acquired pneumonia. JK Sci. 2006;8(2):79-82.
- Capoor MR, Nair D, Aggarwal P, et al. Rapid diagnosis of community-acquired pneumonia using the BacT/Alert 3D system. Braz J Infect Dis. 2006;10(5):352-6.
- Indian Society of Nephrology Vaccination Work Group. Guidelines for vaccination in chronic kidney disease. Indian J Nephrol. 2016;26(Suppl 1):S1-30. Available at: http://isn-india.org/images/Indian-Society-of-Nephrology-Guidelines-for-vaccination-of-Chronic-Kidney-Disease.pdf. Accessed: 12 Aug 2021.

- Wankhedkar R, Tandon RN, Monga VK, et al. Life course immunization guidebook: a quick reference guide. Indian Medical Association; December 2018. Available from: https://www.ima-india.org/ima/pdfdata/IMA\_LifeCourse\_Immunization\_Guide\_2018\_DEC21.pdf. Accessed: 27 Sep 2021.
- Dhar R, Ghoshal AG, Guleria R, et al. Clinical practice guidelines 2019: Indian consensus-based recommendations on pneumococcal vaccination for adults. Lung India. 2020;37(Suppl):S19-29.
- Koul PA, Swaminathan S, Rajgopal T, et al. Adult immunization in occupational settings: a consensus of Indian experts. Indian J Occup Environ Med. 2020;24(1):3-15.
- Geno KA, Gilbert GL, Song JY, et al. Pneumococcal capsules and their types: past, present, and future. Clin Microbiol Rev. 2015;28(3):871-99.
- Hausdorff WP, Hanage WP. Interim results of an ecological experiment conjugate vaccination against the pneumococcus and serotype replacement. Hum Vaccin Immunother. 2016;12(2):358-74.
- AlonsoDeVelasco E, Verheul AFM, Verhoef J, et al. *Streptococcus pneumoniae*: virulence factors, pathogenesis, and vaccines. Microbiol Rev. 1995;59(4):591-603.
- Prevention of pneumococcal disease: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 1997;46(RR-8):1-24.
- Austrian R. A brief history of pneumococcal vaccines. Drugs Aging. 1999;15(Suppl 1):1-10.
- Shapiro ED, Berg AT, Austrian R, et al. The protective efficacy of polyvalent pneumococcal polysaccharide vaccine. N Engl J Med. 1991;325(21):1453-60.
- Stein KE. Thymus-independent and thymus-dependent responses to polysaccharide antigens. J Infect Dis. 1992;165(Suppl 1):S49-52.
- Borrow R, Health PT, Siegrist CA. Use of pneumococcal polysaccharide vaccine in children: what is the evidence? Curr Opin Infect Dis. 2012;25(3):292-303.
- Jackson LA, Neuzil KM, Yu O, et al. Effectiveness of pneumococcal polysaccharide vaccine in older adults. N Engl J Med. 2003;348(18):1747-55.

- Leventer-Roberts M, Feldman BS, Brufman I, et al. Effectiveness of 23-valent pneumococcal polysaccharide vaccine against invasive disease and hospital-treated pneumonia among people aged ≥65 years: a retrospective case-control study. Clin Infect Dis. 2015;60(10):1472-80.
- Wright PF, Sell SH, Vaughn WK, et al. Clinical studies of pneumococcal vaccines in infants. II. Efficacy and effect on nasopharyngeal carriage. Rev Infect Dis. 1981;3(Suppl):S108-12.
- Torres A, Bonanni P, Hryniewicz W, et al. Pneumococcal vaccination: what have we learnt so far and what can we expect in the future? Eur J Clin Microbiol Infect Dis. 2015;34(1):19-31.
- Nuorti JP, Whitney CG, Centers for Disease Control and Prevention. Prevention of pneumococcal disease among infants and children use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2010;59(RR-11):1-18.
- <sup>28</sup> Reinert RR, Paradiso P, Fritzell B. Advances in pneumococcal vaccines: the 13-valent pneumococcal conjugate vaccine received market authorization in Europe. Expert Rev Vaccines. 2010;9(3):229-36.
- Bonten MJM, Huijts SM, Bolkenbaas M, et al. Polysaccharide conjugate vaccine against pneumococcal pneumonia in adults. N Engl J Med. 2015;372(12):1114-25.
- McLaughlin JM, Jiang Q, Isturiz RE, et al. Effectiveness of 13-valent pneumococcal conjugate vaccine against hospitalization for community-acquired pneumonia in older US adults: a test-negative design. Clin Infect Dis. 2018;67(10):1498-506.
- US Food and Drug Administration. Guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. Rockville, MD: Center for Biologics Evaluation and Research; September 2007.

# **Document Approval Record**

**Document Name:** B1851214 Clinical Protocol, 15 Oct 2021

Document Title: A PHASE 4, OPEN-LABEL, SINGLE-ARM, MULTICENTER STUDY T

O DESCRIBE THE SAFETY OF 13-VALENT PNEUMOCOCCAL CON

JUGATE

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|------------------|
| PPD | 15-Oct-2021 18 05 23 | Final Approval |
| PPD | 15-Oct-2021 19 17 09 | Final Approval |